CLINICAL TRIAL: NCT00779766
Title: Efficacy, Immunogenicity and Safety of GlaxoSmithKline Biologicals' HPV GSK 580299 Vaccine in Healthy Chinese Female Subjects
Brief Title: Efficacy, Immunogenicity and Safety of GSK Biologicals' HPV GSK 580299 Vaccine in Healthy Chinese Female Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 107638
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2019-06-10 (Actual); Status verified 2019-05

CONDITIONS: Infections, Papillomavirus
Keywords: Human papillomavirus; vaccine; cervical cancer; cervical infection
MeSH Terms: conditions — Papillomavirus Infections; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Cervarix Group (Experimental): Subjects received 3 doses of Cervarix™ vaccine. Cervarix™ vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: HPV GSK 580299 vaccine
- Placebo Group (Placebo Comparator): Subjects received 3 doses of placebo. Placebo was administered intramuscularly in the deltoid muscle of the non-dominant arm according to a 0, 1, 6-month schedule.
  Interventions: Biological: Placebo control

INTERVENTIONS:
Biological: HPV GSK 580299 vaccine — Subjects were planned to receive three doses of the study vaccine administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: Cervarix Group
Biological: Placebo control — Subjects were planned to receive three doses of the placebo control administered intramuscularly according to a 0, 1, 6 month vaccination schedule.
  Arms: Placebo Group

SUMMARY:
This is a multicenter study in which women are planned to receive either the HPV vaccine or control. Study participation will last approximately 72 months and involves a total of thirteen or fourteen scheduled visits.

Originally, the study was planned for 24 months. It was then extended for 2 more years with 4 additional visits (study end at Month 48).

The protocol posting has been updated as the study was extended by additional 2 years with two or three additional visits (study end at Month 72) for subjects who consent to participate in the extension.

DETAILED DESCRIPTION:
This protocol posting has been updated following protocol amendment 6 dated 24 April 2014.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese females between and including 18 and 25 years of age at the time of the first vaccination.
* Subjects who the investigator believes that they can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to enrolment.
* Healthy subjects as established by medical history and history-directed clinical examination before entering into the study.
* Subjects must not be pregnant. Absence of pregnancy will be verified with a urine pregnancy test.
* Subjects must be of non-childbearing potential, or if of childbearing potential, they must be abstinent or have practiced adequate contraception for 30 days prior to vaccination and agree to continue such precautions for 2 months after completion of the vaccination series.
* Subject must have one single intact cervix.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days before and 30 days after (i.e., Days 0-29) the first dose of vaccine.
* Concurrently participating in another clinical study, at any time during the study period (up to Month 24), in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* A subject planning to become pregnant, likely to become pregnant (as determined by the investigator) or planning to discontinue contraceptive precautions during the study period and up to two months after the last vaccine dose.
* Pregnant or breastfeeding. Subjects must be at least three months post-pregnancy and not breastfeeding to enter the study.
* Previous vaccination against HPV or planned administration of any HPV vaccine other than that foreseen by the protocol during the study period.
* Previous administration of components of the investigational vaccine.
* History of chronic condition(s) requiring treatment such as cancer or autoimmune disease.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the vaccine.
* Hypersensitivity to latex.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of having had colposcopy or has planned a colposcopy to evaluate an abnormal cervical cytology (Pap smear) test.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6081 (Actual)
Dates: Start 2008-10-22 (Actual); Primary Completion 2011-09-06 (Actual); Study Completion 2016-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- China (4):
  - GSK Investigational Site, Jintan, Jiangsu
  - GSK Investigational Site, Lianshui, Jiangsu
  - GSK Investigational Site, Xuzhou, Jiangsu
  - GSK Investigational Site, Yancheng, Jiangsu

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Background] Zhao FH, Zhu FC, Chen W, Li J, Hu YM, Hong Y, Zhang YJ, Pan QJ, Zhu JH, Zhang X, Chen Y, Tang H, Zhang H, Durand C, Datta SK, Struyf F, Bi D; HPV-039 study group. Baseline prevalence and type distribution of human papillomavirus in healthy Chinese women aged 18-25 years enrolled in a clinical trial. Int J Cancer. 2014 Dec 1;135(11):2604-11. doi: 10.1002/ijc.28896. Epub 2014 May 20. PMID 24740547
- [Background] Zhu FC, Chen W, Hu YM, Hong Y, Li J, Zhang X, Zhang YJ, Pan QJ, Zhao FH, Yu JX, Zhang YS, Yang X, Zhang CF, Tang H, Zhang H, Lebacq M, David MP, Datta SK, Struyf F, Bi D, Descamps D; HPV-039 study group. Efficacy, immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine in healthy Chinese women aged 18-25 years: results from a randomized controlled trial. Int J Cancer. 2014 Dec 1;135(11):2612-22. doi: 10.1002/ijc.28897. Epub 2014 May 20. PMID 24740596
- [Background] Zhu FC, Hu SY, Hong Y, Hu YM, Zhang X, Zhang YJ, Pan QJ, Zhang WH, Zhao FH, Zhang CF, Yang X, Yu JX, Zhu J, Zhu Y, Chen F, Zhang Q, Wang H, Wang C, Bi J, Xue S, Shen L, Zhang YS, He Y, Tang H, Karkada N, Suryakiran P, Bi D, Struyf F. Efficacy, immunogenicity, and safety of the HPV-16/18 AS04-adjuvanted vaccine in Chinese women aged 18-25 years: event-triggered analysis of a randomized controlled trial. Cancer Med. 2017 Jan;6(1):12-25. doi: 10.1002/cam4.869. Epub 2016 Dec 20. PMID 27998015
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- [Derived] Chen S, Du Q, Yin J, Xu X, Chen W, Pan Q, Zhang X, Hong Y, Zhang W, Liu B, Cui J, Hu S, Zhao F. HPV genotyping agreement between paired cervical cytological sample and biopsy across lesion severity and vaccination. Virol J. 2025 Jun 2;22(1):176. doi: 10.1186/s12985-025-02791-x. PMID 40452051
- [Derived] Welby S, Rosillon D, Feng Y, Borys D. Progression from human papillomavirus (HPV) infection to cervical lesion or clearance in women (18-25 years): Natural history study in the control arm subjects of AS04-HPV-16/18 vaccine efficacy study in China between 2008 and 2016. Expert Rev Vaccines. 2022 Mar;21(3):407-413. doi: 10.1080/14760584.2022.2021077. Epub 2022 Jan 24. PMID 34939897
- [Derived] Zhao S, Hu S, Xu X, Zhang X, Pan Q, Chen F, Zhao F. Impact of HPV-16/18 AS04-adjuvanted vaccine on preventing subsequent infection and disease after excision treatment: post-hoc analysis from a randomized controlled trial. BMC Infect Dis. 2020 Nov 16;20(1):846. doi: 10.1186/s12879-020-05560-z. PMID 33198657
- [Derived] Hu S, Xu X, Zhu F, Hong Y, Hu Y, Zhang X, Pan Q, Zhang W, Zhang C, Yang X, Yu J, Zhu J, Zhu Y, Chen F, Zhao S, Karkada N, Tang H, Bi D, Struyf F, Zhao F. Efficacy of the AS04-adjuvanted HPV-16/18 vaccine in young Chinese women with oncogenic HPV infection at baseline: post-hoc analysis of a randomized controlled trial. Hum Vaccin Immunother. 2021 Apr 3;17(4):955-964. doi: 10.1080/21645515.2020.1829411. Epub 2020 Nov 12. PMID 33180670
- [Derived] Hu Y, Zhang X, He Y, Ma Z, Xie Y, Lu X, Xu Y, Zhang Y, Jiang Y, Xiao H, Struyf F, Folschweiller N, Jiang J, Poncelet S, Karkada N, Jastorff A, Borys D. Long-term persistence of immune response to the AS04-adjuvanted HPV-16/18 vaccine in Chinese girls aged 9-17 years: Results from an 8-9-year follow-up phase III open-label study. Asia Pac J Clin Oncol. 2020 Dec;16(6):392-399. doi: 10.1111/ajco.13398. Epub 2020 Aug 11. PMID 32780946
- [Derived] Chen J, Gopala K, Akarsh PK, Struyf F, Rosillon D. Prevalence and Incidence of Human Papillomavirus (HPV) Infection Before and After Pregnancy: Pooled Analysis of the Control Arms of Efficacy Trials of HPV-16/18 AS04-Adjuvanted Vaccine. Open Forum Infect Dis. 2019 Dec 4;6(12):ofz486. doi: 10.1093/ofid/ofz486. eCollection 2019 Dec. PMID 31824976
- [Derived] Zhu FC, Hu SY, Hong Y, Hu YM, Zhang X, Zhang YJ, Pan QJ, Zhang WH, Zhao FH, Zhang CF, Yang X, Yu JX, Zhu J, Zhu Y, Chen F, Zhang Q, Wang H, Wang C, Bi J, Xue S, Shen L, Zhang YS, He Y, Tang H, Karkada N, Suryakiran P, Bi D, Struyf F. Efficacy, immunogenicity and safety of the AS04-HPV-16/18 vaccine in Chinese women aged 18-25 years: End-of-study results from a phase II/III, randomised, controlled trial. Cancer Med. 2019 Oct;8(14):6195-6211. doi: 10.1002/cam4.2399. Epub 2019 Jul 15. PMID 31305011
- [Derived] Zhu F, Li J, Hu Y, Zhang X, Yang X, Zhao H, Wang J, Yang J, Xia G, Dai Q, Tang H, Suryakiran P, Datta SK, Descamps D, Bi D, Struyf F. Immunogenicity and safety of the HPV-16/18 AS04-adjuvanted vaccine in healthy Chinese girls and women aged 9 to 45 years. Hum Vaccin Immunother. 2014;10(7):1795-806. doi: 10.4161/hv.28702. PMID 25424785
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 107638 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This record provides the end-of-study analysis, including analyses at Month 24, 48, 57 and 72.
Pre-assignment Details: Out of the 6081 subjects enrolled, 2 did not have any subject or vaccine number allocated and 28 did not receive any study vaccine dose, hence only 6051 subjects started the study.
Groups:
- Cervarix Group: Subjects received 3 doses of Cervarix vaccine. Cervarix vaccine was administered intramuscularly in the deltoid muscle of the non-dominant arm according to a 0, 1, 6-month schedule.
Period: Month 24
Arm/Group | Cervarix Group | Placebo Group
Started | 3026 | 3025
Completed | 2694 | 2693
Not Completed | 332 | 332
Not completed — Serious Adverse Event | 2 | 3
Not completed — Adverse Event | 3 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 159 | 127
Not completed — Migrated/moved from study area | 138 | 162
Not completed — Lost to Follow-up | 9 | 9
Not completed — Other | 18 | 27
Period: Month 48
Arm/Group | Cervarix Group | Placebo Group
Started | 2703 | 2727
Completed | 2529 | 2559
Not Completed | 174 | 168
Not completed — Withdrawal by Subject | 68 | 63
Not completed — Migrated/moved from study area | 76 | 75
Not completed — Lost to Follow-up | 29 | 30
Not completed — Other | 1 | 0
Period: Month 72
Arm/Group | Cervarix Group | Placebo Group
Started | 2319 | 2347
Completed | 2134 | 2158
Not Completed | 185 | 189
Not completed — Withdrawal by Subject | 55 | 71
Not completed — Migrated/moved from study area | 124 | 109
Not completed — Lost to Follow-up | 6 | 8
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix Group | Placebo Group | Total
Number analyzed (Participants) | 3026 | 3025 | 6051
Age, Continuous [Mean (Standard Deviation); unit: Years] | 23.0 (1.70) | 23.0 (1.75) | 23.0 (1.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3026 | 3025 | 6051
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - Chinese Heritage | 3026 | 3025 | 6051

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN1+) and/or Persistent Infection (6 Month+ Definition) Associated With Human Papillomavirus (HPV)-16 and/or HPV-18 at Month 24
Description: CIN1+ = CIN 1, 2, and 3, low/high-grade cervical glandular intraepithelial neoplasia (L/HCGIN), adenocarcinoma in-situ (AIS) or invasive cervical cancer. Persistent infection (6-month+ definition) = at least 2 positive HPV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assays for the same viral genotype with no negative DNA sample between the 2 positive DNA samples, over an interval of approximately 6 months. The analyses were done on subjects HPV DNA negative at baseline (Month 0) and Month 6 and seronegative at baseline (Month 0) or on subjects DNA negative at baseline (Month 0) and Month 6, regardless of initial serostatus.
Time Frame: At Month 24
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for efficacy, which included all evaluable subjects for whom efficacy data were available and who had a normal or low-grade cytology (negative or atypical squamous cells of undetermined significance (ASC-US) or low-grade squamous intraepithelial lesion (LSIL)) at Month 0.
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2775 | 2764
Subjects
  Sero negative, DNA negative HPV-16/18: number analyzed (Participants) | 2497 | 2502
  Sero negative, DNA negative HPV-16/18 | 1 | 17
  Sero negative, DNA negative HPV-16: number analyzed (Participants) | 1937 | 1884
  Sero negative, DNA negative HPV-16 | 1 | 15
  Sero negative, DNA negative HPV-18: number analyzed (Participants) | 2320 | 2314
  Sero negative, DNA negative HPV-18 | 0 | 3
  DNA negative, HPV-16/18 | 1 | 27
  DNA negative, HPV-16: number analyzed (Participants) | 2677 | 2672
  DNA negative, HPV-16 | 1 | 21
  DNA negative, HPV-18: number analyzed (Participants) | 2738 | 2731
  DNA negative, HPV-18 | 0 | 7

2. Primary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN1+) and/or Persistent Infection (6 Month+ Definition) Associated With Human Papillomavirus (HPV)-16 and/or HPV-18 at Month 48
Description: as for outcome 1
Time Frame: At Month 48
Population: The analysis was performed on the ATP cohort for efficacy, which included all evaluable subjects for whom data concerning efficacy outcome measures were available and who had a normal or low-grade cytology (negative or ASC-US or LSIL) at Month 0.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2803 | 2799
Participants
  Sero negative, DNA negative HPV-16/18: number analyzed (Participants) | 2522 | 2531
  Sero negative, DNA negative HPV-16/18 | 2 | 45
  Sero negative, DNA negative HPV-16: number analyzed (Participants) | 1958 | 1908
  Sero negative, DNA negative HPV-16 | 2 | 33
  Sero negative, DNA negative HPV-18: number analyzed (Participants) | 2320 | 2314
  Sero negative, DNA negative HPV-18 | 0 | 14
  DNA negative, HPV-16/18 | 2 | 61
  DNA negative, HPV-16: number analyzed (Participants) | 2705 | 2707
  DNA negative, HPV-16 | 2 | 45
  DNA negative, HPV-18: number analyzed (Participants) | 2766 | 2765
  DNA negative, HPV-18 | 0 | 18

3. Primary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN1+) and/or Persistent Infection (6 Month+ Definition) Associated With Human Papillomavirus (HPV)-16 and/or HPV-18 at Month 57
Description: as for outcome 1
Time Frame: At Month 57
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2805 | 2802
Participants
  Sero negative, DNA negative HPV-16/18: number analyzed (Participants) | 2524 | 2535
  Sero negative, DNA negative HPV-16/18 | 2 | 60
  Sero negative, DNA negative HPV-16: number analyzed (Participants) | 1959 | 1909
  Sero negative, DNA negative HPV-16 | 2 | 43
  Sero negative, DNA negative HPV-18: number analyzed (Participants) | 2346 | 2344
  Sero negative, DNA negative HPV-18 | 0 | 19
  DNA negative HPV-16/18 | 2 | 78
  DNA negative HPV-16: number analyzed (Participants) | 2707 | 2710
  DNA negative HPV-16 | 2 | 57
  DNA negative HPV-18: number analyzed (Participants) | 2768 | 2768
  DNA negative HPV-18 | 0 | 23

4. Primary Outcome: Number of Subjects With Histopathologically-confirmed Cervical Intraepithelial Neoplasia (CIN1+) and/or Persistent Infection (6 Month+ Definition) Associated With Human Papillomavirus (HPV)-16 and/or HPV-18 at Month 72
Description: as for outcome 1
Time Frame: At Month 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2804 | 2801
Participants
  Sero negative, DNA negative HPV-16/18: number analyzed (Participants) | 2523 | 2534
  Sero negative, DNA negative HPV-16/18 | 2 | 69
  Sero negative, DNA negative HPV-16: number analyzed (Participants) | 1958 | 1908
  Sero negative, DNA negative HPV-16 | 2 | 50
  Sero negative, DNA negative HPV-18: number analyzed (Participants) | 2345 | 2344
  Sero negative, DNA negative HPV-18 | 0 | 21
  DNA negative HPV-16/18 | 2 | 91
  DNA negative HPV-16: number analyzed (Participants) | 2706 | 2709
  DNA negative HPV-16 | 2 | 68
  DNA negative HPV-18: number analyzed (Participants) | 2767 | 2767
  DNA negative HPV-18 | 0 | 26

5. Secondary Outcome: Number of Subjects With Incident Cervical Infection With HPV-16 and/or HPV-18
Description: HPV-16 and/or HPV-18 incident infection is defined as at least one positive HPV-16 or HPV-18 DNA PCR assay at the time point considered. - DNA- and sero-: subjects HPV DNA negative at Months 0 and 6 by PCR and seronegative at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA) - Overall: subjects DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus.
Time Frame: At Months 24,48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2807 | 2802
Participants
  Sero negative, DNA negative HPV-16/18 M24: number analyzed (Participants) | 2497 | 2502
  Sero negative, DNA negative HPV-16/18 M24 | 15 | 49
  Sero negative, DNA negative HPV-16 M24: number analyzed (Participants) | 1935 | 1884
  Sero negative, DNA negative HPV-16 M24 | 9 | 30
  Sero negative, DNA negative HPV-18 M24: number analyzed (Participants) | 2321 | 2314
  Sero negative, DNA negative HPV-18 M24 | 7 | 21
  DNA negative HPV-16/18 M24: number analyzed (Participants) | 2776 | 2764
  DNA negative HPV-16/18 M24 | 20 | 70
  DNA negative HPV-16 M24: number analyzed (Participants) | 2677 | 2672
  DNA negative HPV-16 M24 | 13 | 43
  DNA negative HPV-18 M24: number analyzed (Participants) | 2740 | 2731
  DNA negative HPV-18 M24 | 8 | 30
  Sero negative, DNA negative HPV-16/18 M48: number analyzed (Participants) | 2519 | 2527
  Sero negative, DNA negative HPV-16/18 M48 | 22 | 96
  Sero negative, DNA negative HPV-16 M48: number analyzed (Participants) | 1953 | 1905
  Sero negative, DNA negative HPV-16 M48 | 13 | 62
  Sero negative, DNA negative HPV-18 M48: number analyzed (Participants) | 2341 | 2337
  Sero negative, DNA negative HPV-18 M48 | 10 | 39
  DNA negative HPV-16/18 M48: number analyzed (Participants) | 2397 | 2424
  DNA negative HPV-16/18 M48 | 1 | 21
  DNA negative HPV-18 M48: number analyzed (Participants) | 2230 | 2241
  DNA negative HPV-18 M48 | 0 | 5
  DNA negative HPV-16 M48: number analyzed (Participants) | 1859 | 1830
  DNA negative HPV-16 M48 | 1 | 16
  Sero negative, DNA negative HPV-16/18 M57: number analyzed (Participants) | 2525 | 2535
  Sero negative, DNA negative HPV-16/18 M57 | 29 | 142
  Sero negative, DNA negative HPV-16 M57: number analyzed (Participants) | 1958 | 1909
  Sero negative, DNA negative HPV-16 M57 | 16 | 92
  Sero negative, DNA negative HPV-18 M57: number analyzed (Participants) | 2347 | 2344
  Sero negative, DNA negative HPV-18 M57 | 14 | 57
  DNA negative HPV-16/18 M57 | 43 | 189
  DNA negative HPV-16 M57: number analyzed (Participants) | 2708 | 2710
  DNA negative HPV-16 M57 | 26 | 127
  DNA negative HPV-18 M57: number analyzed (Participants) | 2770 | 2768
  DNA negative HPV-18 M57 | 18 | 74
  Sero negative, DNA negative HPV-16/18 M72: number analyzed (Participants) | 2524 | 2534
  Sero negative, DNA negative HPV-16/18 M72 | 34 | 156
  Sero negative, DNA negative HPV-16 M72: number analyzed (Participants) | 1957 | 1908
  Sero negative, DNA negative HPV-16 M72 | 21 | 103
  Sero negative, DNA negative HPV-18 M72: number analyzed (Participants) | 2346 | 2344
  Sero negative, DNA negative HPV-18 M72 | 14 | 63
  DNA negative HPV-16/18 M72: number analyzed (Participants) | 1806 | 2801
  DNA negative HPV-16/18 M72 | 49 | 204
  DNA negative HPV-16 M72: number analyzed (Participants) | 2707 | 2709
  DNA negative HPV-16 M72 | 32 | 139
  DNA negative HPV-18 M72: number analyzed (Participants) | 2769 | 2767
  DNA negative HPV-18 M72 | 18 | 81

6. Secondary Outcome: Number of Subjects With Persistent Cervical Infection (6-month+ Definition) With HPV-16 and/or HPV-18
Description: Persistent HPV-16 and/or HPV-18 infection (6-month+ definition) = at least 2 positive HPV deoxyribonucleic acid (DNA) polymerase chain reaction (PCR) assays for the same viral genotype with no negative DNA sample between the two positive DNA samples, over an interval of approximately 6 months. Subjects had at least 5 months of follow-up after Month 12. DNA- and sero-: subjects HPV DNA negative at Months 0 and 6 by PCR and seronegative at Month 0 for the corresponding HPV-type by ELISA Overall: subjects DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2762 | 2748
Participants
  Sero negative, DNA negative HPV-16/18 M24: number analyzed (Participants) | 2332 | 2326
  Sero negative, DNA negative HPV-16/18 M24 | 1 | 15
  Sero negative, DNA negative HPV-16 M24: number analyzed (Participants) | 1810 | 1747
  Sero negative, DNA negative HPV-16 M24 | 1 | 13
  Sero negative, DNA negative HPV-18 M24: number analyzed (Participants) | 2168 | 2154
  Sero negative, DNA negative HPV-18 M24 | 0 | 3
  Overall HPV-16/18 M24: number analyzed (Participants) | 2596 | 2569
  Overall HPV-16/18 M24 | 1 | 24
  Overall HPV-16 M24: number analyzed (Participants) | 2509 | 2488
  Overall HPV-16 M24 | 1 | 18
  Overall HPV-18 M24: number analyzed (Participants) | 2565 | 2537
  Overall HPV-18 M24 | 0 | 7
  Sero negative, DNA negative HPV-16/18 M48: number analyzed (Participants) | 2464 | 2474
  Sero negative, DNA negative HPV-16/18 M48 | 2 | 39
  Sero negative, DNA negative HPV-16 M48: number analyzed (Participants) | 1915 | 1864
  Sero negative, DNA negative HPV-16 M48 | 2 | 30
  Sero negative, DNA negative HPV-18 M48: number analyzed (Participants) | 2290 | 2288
  Sero negative, DNA negative HPV-18 M48 | 0 | 11
  Overall HPV-16/18 M48: number analyzed (Participants) | 2742 | 2728
  Overall HPV-16/18 M48 | 2 | 53
  Overall HPV-16 M48: number analyzed (Participants) | 2647 | 2639
  Overall HPV-16 M48 | 2 | 40
  Overall HPV-18 M48: number analyzed (Participants) | 2706 | 2694
  Overall HPV-18 M48 | 0 | 15
  Sero negative, DNA negative HPV-16/18 M57: number analyzed (Participants) | 2480 | 2488
  Sero negative, DNA negative HPV-16/18 M57 | 2 | 54
  Sero negative, DNA negative HPV-16 M57: number analyzed (Participants) | 1928 | 1875
  Sero negative, DNA negative HPV-16 M57 | 2 | 39
  Sero negative, DNA negative HPV-18 M57: number analyzed (Participants) | 2306 | 2298
  Sero negative, DNA negative HPV-18 M57 | 0 | 17
  Overall HPV-16/18 M57: number analyzed (Participants) | 2759 | 2744
  Overall HPV-16/18 M57 | 2 | 70
  Overall HPV-16 M57: number analyzed (Participants) | 2663 | 2655
  Overall HPV-16 M57 | 2 | 51
  Overall HPV-18 M57: number analyzed (Participants) | 2723 | 2710
  Overall HPV-18 M57 | 0 | 21
  Sero negative, DNA negative HPV-16/18 M72: number analyzed (Participants) | 2483 | 2492
  Sero negative, DNA negative HPV-16/18 M72 | 2 | 63
  Sero negative, DNA negative HPV-16 M72: number analyzed (Participants) | 1929 | 1876
  Sero negative, DNA negative HPV-16 M72 | 2 | 46
  Sero negative, DNA negative HPV-18 M72: number analyzed (Participants) | 2309 | 2303
  Sero negative, DNA negative HPV-18 M72 | 0 | 19
  Overall HPV-16/18 M72 | 2 | 83
  Overall HPV-16 M72: number analyzed (Participants) | 2666 | 2659
  Overall HPV-16 M72 | 2 | 62
  Overall HPV-18 M72: number analyzed (Participants) | 2726 | 2714
  Overall HPV-18 M72 | 0 | 24

7. Secondary Outcome: Number of Subjects With Persistent Cervical Infection (12-month+ Definition) With HPV-16 and/or HPV-18
Description: Persistent infection (12-month+ definition) is defined as the detection of the same HPV type(s) (by PCR) in cervical samples at all available time points over an interval of approximately 12 months. Subjects had at least 10 months of follow-up after Month 12. DNA- and sero-: subjects HPV DNA negative at Months 0 and 6 by PCR and seronegative at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA). Overall: subjects DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2702 | 2709
Subjects
  Sero negative, DNA negative HPV-16/18 M24: number analyzed (Participants) | 1111 | 1091
  Sero negative, DNA negative HPV-16/18 M24 | 0 | 2
  Sero negative, DNA negative HPV-16 M24: number analyzed (Participants) | 799 | 768
  Sero negative, DNA negative HPV-16 M24 | 0 | 2
  Sero negative, DNA negative HPV-18 M24: number analyzed (Participants) | 1034 | 1014
  Sero negative, DNA negative HPV-18 M24 | 0 | 0
  Overall, HPV-16/18 M24: number analyzed (Participants) | 1304 | 1257
  Overall, HPV-16/18 M24 | 0 | 2
  Overall, HPV-16 M24: number analyzed (Participants) | 1261 | 1216
  Overall, HPV-16 M24 | 0 | 2
  Overall, HPV-18 M24: number analyzed (Participants) | 1285 | 1242
  Overall, HPV-18 M24 | 0 | 0
  Sero negative, DNA negative HPV-16/18 M48: number analyzed (Participants) | 2397 | 2424
  Sero negative, DNA negative HPV-16/18 M48 | 1 | 21
  Sero negative, DNA negative HPV-16 M48: number analyzed (Participants) | 1859 | 1830
  Sero negative, DNA negative HPV-16 M48 | 1 | 16
  Sero negative, DNA negative HPV-18 M48: number analyzed (Participants) | 2230 | 2241
  Sero negative, DNA negative HPV-18 M48 | 0 | 5
  Overall, HPV-16/18 M48: number analyzed (Participants) | 2668 | 2673
  Overall, HPV-16/18 M48 | 1 | 22
  Overall, HPV-16 M48: number analyzed (Participants) | 2575 | 2587
  Overall, HPV-16 M48 | 1 | 17
  Overall, HPV-18 M48: number analyzed (Participants) | 2633 | 2639
  Overall, HPV-18 M48 | 0 | 5
  Sero negative, DNA negative HPV-16/18 M57: number analyzed (Participants) | 2425 | 2455
  Sero negative, DNA negative HPV-16/18 M57 | 1 | 32
  Sero negative, DNA negative HPV-16 M57: number analyzed (Participants) | 1880 | 1856
  Sero negative, DNA negative HPV-16 M57 | 1 | 24
  Sero negative, DNA negative HPV-18 M57: number analyzed (Participants) | 2257 | 2269
  Sero negative, DNA negative HPV-18 M57 | 0 | 8
  Overall, HPV-16/18 M57: number analyzed (Participants) | 2699 | 2706
  Overall, HPV-16/18 M57 | 1 | 37
  Overall, HPV-16 M57: number analyzed (Participants) | 2604 | 2620
  Overall, HPV-16 M57 | 1 | 29
  Overall, HPV-18 M57: number analyzed (Participants) | 2664 | 2672
  Overall, HPV-18 M57 | 0 | 8
  Sero negative, DNA negative HPV-16/18 M72: number analyzed (Participants) | 2428 | 2458
  Sero negative, DNA negative HPV-16/18 M72 | 1 | 32
  Sero negative, DNA negative HPV-16 M72: number analyzed (Participants) | 1882 | 1857
  Sero negative, DNA negative HPV-16 M72 | 1 | 24
  Sero negative, DNA negative HPV-18 M72: number analyzed (Participants) | 2258 | 2273
  Sero negative, DNA negative HPV-18 M72 | 0 | 8
  Overall, HPV-16/18 M72 | 1 | 38
  Overall, HPV-16 M72: number analyzed (Participants) | 2607 | 2622
  Overall, HPV-16 M72 | 1 | 30
  Overall, HPV-18 M72: number analyzed (Participants) | 2666 | 2675
  Overall, HPV-18 M72 | 0 | 8

8. Secondary Outcome: Number of Subjects With Incident Cervical Infection With Any Oncogenic HPV Type
Description: Oncogenic HPV types assessed were HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68 individually or in combination. Subjects were HPV DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus. HRW-HPV=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HR-HPV=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2812 | 2812
Subjects
  HPV-16 M24: number analyzed (Participants) | 2677 | 2672
  HPV-16 M24 | 13 | 43
  HPV-18 M24: number analyzed (Participants) | 2740 | 2731
  HPV-18 M24 | 8 | 30
  HPV-31 M24: number analyzed (Participants) | 2745 | 2733
  HPV-31 M24 | 14 | 25
  HPV-33 M24: number analyzed (Participants) | 2738 | 2733
  HPV-33 M24 | 19 | 22
  HPV-35 M24: number analyzed (Participants) | 2764 | 2753
  HPV-35 M24 | 17 | 15
  HPV-39 M24: number analyzed (Participants) | 2716 | 2723
  HPV-39 M24 | 42 | 32
  HPV-45 M24: number analyzed (Participants) | 2751 | 2751
  HPV-45 M24 | 8 | 17
  HPV-51 M24: number analyzed (Participants) | 2712 | 2708
  HPV-51 M24 | 69 | 57
  HPV-52 M24: number analyzed (Participants) | 2626 | 2615
  HPV-52 M24 | 90 | 87
  HPV-56 M24: number analyzed (Participants) | 2741 | 2730
  HPV-56 M24 | 34 | 37
  HPV-58 M24: number analyzed (Participants) | 2730 | 2718
  HPV-58 M24 | 28 | 34
  HPV-59 M24: number analyzed (Participants) | 2771 | 2746
  HPV-59 M24 | 16 | 20
  HPV-66 M24: number analyzed (Participants) | 2737 | 2715
  HPV-66 M24 | 37 | 33
  HPV-68 M24: number analyzed (Participants) | 2732 | 2734
  HPV-68 M24 | 33 | 32
  HPV-31/33/45 M24: number analyzed (Participants) | 2780 | 2773
  HPV-31/33/45 M24 | 36 | 60
  HPV-16/18/31/33/45 M24: number analyzed (Participants) | 2780 | 2774
  HPV-16/18/31/33/45 M24 | 54 | 126
  HRW-HPV M24: number analyzed (Participants) | 2780 | 2774
  HRW-HPV M24 | 313 | 324
  HR-HPV M24: number analyzed (Participants) | 2780 | 2774
  HR-HPV M24 | 323 | 364
  HPV-16 M48: number analyzed (Participants) | 2702 | 2702
  HPV-16 M48 | 18 | 88
  HPV-18 M48: number analyzed (Participants) | 2764 | 2760
  HPV-18 M48 | 13 | 50
  HPV-31 M48: number analyzed (Participants) | 2770 | 2762
  HPV-31 M48 | 29 | 59
  HPV-33 M48: number analyzed (Participants) | 2763 | 2763
  HPV-33 M48 | 29 | 52
  HPV-35 M48: number analyzed (Participants) | 2789 | 2783
  HPV-35 M48 | 35 | 38
  HPV-39 M48: number analyzed (Participants) | 2742 | 2752
  HPV-39 M48 | 80 | 78
  HPV-45 M48: number analyzed (Participants) | 2777 | 2781
  HPV-45 M48 | 13 | 25
  HPV-51 M48: number analyzed (Participants) | 2736 | 2736
  HPV-51 M48 | 117 | 131
  HPV-52 M48: number analyzed (Participants) | 2650 | 2644
  HPV-52 M48 | 168 | 176
  HPV-56 M48: number analyzed (Participants) | 2766 | 2760
  HPV-56 M48 | 63 | 70
  HPV-58 M48: number analyzed (Participants) | 2755 | 2748
  HPV-58 M48 | 56 | 62
  HPV-59 M48: number analyzed (Participants) | 2797 | 2776
  HPV-59 M48 | 35 | 44
  HPV-66 M48: number analyzed (Participants) | 2763 | 2745
  HPV-66 M48 | 74 | 73
  HPV-68 M48: number analyzed (Participants) | 2758 | 2764
  HPV-68 M48 | 59 | 61
  HPV-31/33/45 M48: number analyzed (Participants) | 2806 | 2803
  HPV-31/33/45 M48 | 62 | 119
  HPV-16/18/31/33/45 M48: number analyzed (Participants) | 2806 | 2804
  HPV-16/18/31/33/45 M48 | 89 | 239
  HRW-HPV M48: number analyzed (Participants) | 2806 | 2804
  HRW-HPV M48 | 536 | 591
  HR-HPV M48: number analyzed (Participants) | 2806 | 2804
  HR-HPV M48 | 552 | 646
  HPV-16 M57: number analyzed (Participants) | 2708 | 2710
  HPV-16 M57 | 26 | 127
  HPV-18 M57: number analyzed (Participants) | 2770 | 2768
  HPV-18 M57 | 18 | 74
  HPV-31 M57: number analyzed (Participants) | 2776 | 2770
  HPV-31 M57 | 33 | 74
  HPV-33 M57: number analyzed (Participants) | 2769 | 2771
  HPV-33 M57 | 40 | 69
  HPV-35 M57: number analyzed (Participants) | 2795 | 2791
  HPV-35 M57 | 49 | 55
  HPV-39 M57: number analyzed (Participants) | 2748 | 2760
  HPV-39 M57 | 136 | 121
  HPV-45 M57: number analyzed (Participants) | 2783 | 2789
  HPV-45 M57 | 18 | 38
  HPV-51 M57: number analyzed (Participants) | 2742 | 2743
  HPV-51 M57 | 152 | 187
  HPV-52 M57: number analyzed (Participants) | 2656 | 2652
  HPV-52 M57 | 227 | 264
  HPV-56 M57: number analyzed (Participants) | 2772 | 2767
  HPV-56 M57 | 93 | 106
  HPV-58 M57: number analyzed (Participants) | 2761 | 2756
  HPV-58 M57 | 77 | 99
  HPV-59 M57: number analyzed (Participants) | 2806 | 2784
  HPV-59 M57 | 47 | 62
  HPV-66 M57: number analyzed (Participants) | 2769 | 2752
  HPV-66 M57 | 96 | 111
  HPV-68 M57: number analyzed (Participants) | 2764 | 2772
  HPV-68 M57 | 91 | 95
  HPV-31/33/45 M57: number analyzed (Participants) | 2812 | 2811
  HPV-31/33/45 M57 | 80 | 159
  HPV-16/18/31/33/45 M57 | 120 | 329
  HRW-HPV M57 | 692 | 800
  HR-HPV M57 | 710 | 862
  HPV-16 M72: number analyzed (Participants) | 2707 | 2709
  HPV-16 M72 | 32 | 139
  HPV-18 M72: number analyzed (Participants) | 2769 | 2768
  HPV-18 M72 | 18 | 81
  HPV-31 M72: number analyzed (Participants) | 2775 | 2769
  HPV-31 M72 | 35 | 86
  HPV-33 M72: number analyzed (Participants) | 2768 | 2770
  HPV-33 M72 | 43 | 75
  HPV-35 M72: number analyzed (Participants) | 2794 | 2790
  HPV-35 M72 | 53 | 65
  HPV-39 M72: number analyzed (Participants) | 2747 | 2759
  HPV-39 M72 | 154 | 133
  HPV-45 M72: number analyzed (Participants) | 2782 | 2788
  HPV-45 M72 | 18 | 40
  HPV-51 M72: number analyzed (Participants) | 2741 | 2742
  HPV-51 M72 | 166 | 204
  HPV-52 M72: number analyzed (Participants) | 2655 | 2651
  HPV-52 M72 | 251 | 284
  HPV-56 M72: number analyzed (Participants) | 2771 | 2766
  HPV-56 M72 | 104 | 113
  HPV-58 M72: number analyzed (Participants) | 2760 | 2755
  HPV-58 M72 | 83 | 111
  HPV-59 M72: number analyzed (Participants) | 2802 | 2783
  HPV-59 M72 | 52 | 65
  HPV-66 M72: number analyzed (Participants) | 2768 | 2751
  HPV-66 M72 | 103 | 124
  HPV-68 M72: number analyzed (Participants) | 2763 | 2771
  HPV-68 M72 | 101 | 107
  HPV-31/33/45 M72: number analyzed (Participants) | 2811 | 2810
  HPV-31/33/45 M72 | 85 | 175
  HPV-16/18/31/33/45 M72: number analyzed (Participants) | 2811 | 2811
  HPV-16/18/31/33/45 M72 | 131 | 356
  HRW-HPV M72: number analyzed (Participants) | 2811 | 2811
  HRW-HPV M72 | 744 | 852
  HR-HPV M72: number analyzed (Participants) | 2811 | 2811
  HR-HPV M72 | 764 | 914

9. Secondary Outcome: Number of Subjects With Persistent Cervical Infection (6-month+ Definition) With Any Oncogenic HPV Type
Description: as for outcome 8
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2767 | 2756
Participants
  HPV-16 M24: number analyzed (Participants) | 2509 | 2488
  HPV-16 M24 | 1 | 18
  HPV-18 M24: number analyzed (Participants) | 2565 | 2537
  HPV-18 M24 | 0 | 7
  HPV-31 M24: number analyzed (Participants) | 2568 | 2540
  HPV-31 M24 | 5 | 6
  HPV-33 M24: number analyzed (Participants) | 2562 | 2539
  HPV-33 M24 | 7 | 8
  HPV-35 M24: number analyzed (Participants) | 2585 | 2558
  HPV-35 M24 | 4 | 7
  HPV-39 M24: number analyzed (Participants) | 2540 | 2532
  HPV-39 M24 | 11 | 9
  HPV-45 M24: number analyzed (Participants) | 2573 | 2559
  HPV-45 M24 | 1 | 5
  HPV-51 M24: number analyzed (Participants) | 2544 | 2514
  HPV-51 M24 | 21 | 14
  HPV-52 M24: number analyzed (Participants) | 2466 | 2438
  HPV-52 M24 | 36 | 23
  HPV-56 M24: number analyzed (Participants) | 2566 | 2538
  HPV-56 M24 | 13 | 5
  HPV-58 M24: number analyzed (Participants) | 2553 | 2526
  HPV-58 M24 | 8 | 12
  HPV-59 M24: number analyzed (Participants) | 2591 | 2551
  HPV-59 M24 | 6 | 7
  HPV-66 M24: number analyzed (Participants) | 2564 | 2521
  HPV-66 M24 | 5 | 8
  HPV-68 M24: number analyzed (Participants) | 2558 | 2540
  HPV-68 M24 | 11 | 7
  HPV-31/33/45 M24: number analyzed (Participants) | 2600 | 2576
  HPV-31/33/45 M24 | 12 | 19
  HPV-16/18/31/33/45 M24: number analyzed (Participants) | 2600 | 2577
  HPV-16/18/31/33/45 M24 | 13 | 42
  HRW-HPV M24: number analyzed (Participants) | 2600 | 2577
  HRW-HPV M24 | 114 | 98
  HR-HPV M24: number analyzed (Participants) | 2600 | 2577
  HR-HPV M24 | 115 | 116
  HPV-16 M48: number analyzed (Participants) | 2647 | 2639
  HPV-16 M48 | 2 | 40
  HPV-18 M48: number analyzed (Participants) | 2706 | 2694
  HPV-18 M48 | 0 | 15
  HPV-31 M48: number analyzed (Participants) | 2714 | 2698
  HPV-31 M48 | 10 | 23
  HPV-33 M48: number analyzed (Participants) | 2705 | 2696
  HPV-33 M48 | 12 | 19
  HPV-35 M48: number analyzed (Participants) | 2730 | 2718
  HPV-35 M48 | 13 | 15
  HPV-39 M48: number analyzed (Participants) | 2684 | 2686
  HPV-39 M48 | 34 | 29
  HPV-45 M48: number analyzed (Participants) | 2718 | 2717
  HPV-45 M48 | 7 | 7
  HPV-51 M48: number analyzed (Participants) | 2684 | 2669
  HPV-51 M48 | 49 | 42
  HPV-52 M48: number analyzed (Participants) | 2598 | 2587
  HPV-52 M48 | 84 | 72
  HPV-56 M48: number analyzed (Participants) | 2709 | 2693
  HPV-56 M48 | 25 | 29
  HPV-58 M48: number analyzed (Participants) | 2698 | 2684
  HPV-58 M48 | 25 | 29
  HPV-59 M48: number analyzed (Participants) | 2738 | 2710
  HPV-59 M48 | 14 | 13
  HPV-66 M48: number analyzed (Participants) | 2706 | 2678
  HPV-66 M48 | 19 | 25
  HPV-68 M48: number analyzed (Participants) | 2703 | 2698
  HPV-68 M48 | 21 | 20
  HPV-31/33/45 M48: number analyzed (Participants) | 2747 | 2736
  HPV-31/33/45 M48 | 27 | 46
  HPV-16/18/31/33/45 M48: number analyzed (Participants) | 2747 | 2737
  HPV-16/18/31/33/45 M48 | 29 | 97
  HRW-HPV M48: number analyzed (Participants) | 2747 | 2737
  HRW-HPV M48 | 257 | 275
  HR-HPV M48 | 258 | 312
  HPV-16 M57: number analyzed (Participants) | 2663 | 2655
  HPV-16 M57 | 2 | 51
  HPV-18 M57: number analyzed (Participants) | 2723 | 2710
  HPV-18 M57 | 0 | 21
  HPV-31 M57: number analyzed (Participants) | 2731 | 2714
  HPV-31 M57 | 10 | 29
  HPV-33 M57: number analyzed (Participants) | 2722 | 2712
  HPV-33 M57 | 13 | 25
  HPV-35 M57: number analyzed (Participants) | 2747 | 2734
  HPV-35 M57 | 17 | 18
  HPV-39 M57: number analyzed (Participants) | 2701 | 2702
  HPV-39 M57 | 47 | 41
  HPV-45 M57: number analyzed (Participants) | 2735 | 2733
  HPV-45 M57 | 7 | 8
  HPV-51 M57: number analyzed (Participants) | 2699 | 2685
  HPV-51 M57 | 59 | 58
  HPV-52 M57: number analyzed (Participants) | 2612 | 2602
  HPV-52 M57 | 109 | 97
  HPV-56 M57: number analyzed (Participants) | 2726 | 2709
  HPV-56 M57 | 32 | 36
  HPV-58 M57: number analyzed (Participants) | 2715 | 2699
  HPV-58 M57 | 32 | 40
  HPV-59 M57: number analyzed (Participants) | 2755 | 2726
  HPV-59 M57 | 15 | 15
  HPV-66 M57: number analyzed (Participants) | 2723 | 2694
  HPV-66 M57 | 31 | 29
  HPV-68 M57: number analyzed (Participants) | 2720 | 2714
  HPV-68 M57 | 28 | 30
  HPV-31/33/45 M57: number analyzed (Participants) | 2764 | 2752
  HPV-31/33/45 M57 | 28 | 59
  HPV-16/18/31/33/45 M57: number analyzed (Participants) | 2764 | 2753
  HPV-16/18/31/33/45 M57 | 30 | 126
  HRW-HPV M57: number analyzed (Participants) | 2764 | 2753
  HRW-HPV M57 | 319 | 357
  HR-HPV M57: number analyzed (Participants) | 2764 | 2753
  HR-HPV M57 | 320 | 400
  HPV-16 M72: number analyzed (Participants) | 2666 | 2659
  HPV-16 M72 | 2 | 62
  HPV-18 M72: number analyzed (Participants) | 2726 | 2714
  HPV-18 M72 | 0 | 24
  HPV-31 M72: number analyzed (Participants) | 2734 | 2718
  HPV-31 M72 | 11 | 31
  HPV-33 M72: number analyzed (Participants) | 2725 | 2716
  HPV-33 M72 | 16 | 30
  HPV-35 M72: number analyzed (Participants) | 2750 | 2738
  HPV-35 M72 | 19 | 18
  HPV-39 M72: number analyzed (Participants) | 2703 | 2706
  HPV-39 M72 | 63 | 50
  HPV-45 M72: number analyzed (Participants) | 2738 | 2737
  HPV-45 M72 | 8 | 10
  HPV-51 M72: number analyzed (Participants) | 2702 | 2688
  HPV-51 M72 | 69 | 73
  HPV-52 M72: number analyzed (Participants) | 2614 | 2606
  HPV-52 M72 | 128 | 117
  HPV-56 M72: number analyzed (Participants) | 2728 | 2712
  HPV-56 M72 | 43 | 41
  HPV-58 M72: number analyzed (Participants) | 2718 | 2703
  HPV-58 M72 | 38 | 49
  HPV-59 M72: number analyzed (Participants) | 2758 | 2730
  HPV-59 M72 | 16 | 16
  HPV-66 M72: number analyzed (Participants) | 2726 | 2697
  HPV-66 M72 | 36 | 37
  HPV-68 M72: number analyzed (Participants) | 2723 | 2718
  HPV-68 M72 | 32 | 36
  HPV-31/33/45 M72 | 33 | 68
  HPV-16/18/31/33/45 M72 | 35 | 146
  HRW-HPV M72 | 381 | 418
  HR-HPV M72 | 382 | 466

10. Secondary Outcome: Number of Subjects With Persistent Cervical Infection (12-month+ Definition) With Any Oncogenic HPV Type
Description: as for outcome 8
Time Frame: At Months 24,48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2706 | 2717
Participants
  HPV-16 M24: number analyzed (Participants) | 1261 | 1216
  HPV-16 M24 | 0 | 2
  HPV-18 M24: number analyzed (Participants) | 1285 | 1242
  HPV-18 M24 | 0 | 0
  HPV-31 M24: number analyzed (Participants) | 1283 | 1239
  HPV-31 M24 | 0 | 0
  HPV-33 M24: number analyzed (Participants) | 1287 | 1248
  HPV-33 M24 | 2 | 1
  HPV-35 M24: number analyzed (Participants) | 1298 | 1255
  HPV-35 M24 | 1 | 0
  HPV-39 M24: number analyzed (Participants) | 1272 | 1234
  HPV-39 M24 | 1 | 3
  HPV-45 M24: number analyzed (Participants) | 1292 | 1246
  HPV-45 M24 | 1 | 0
  HPV-51 M24: number analyzed (Participants) | 1281 | 1229
  HPV-51 M24 | 6 | 2
  HPV-52 M24: number analyzed (Participants) | 1240 | 1193
  HPV-52 M24 | 7 | 5
  HPV-56 M24: number analyzed (Participants) | 1283 | 1246
  HPV-56 M24 | 0 | 0
  HPV-58 M24: number analyzed (Participants) | 1273 | 1238
  HPV-58 M24 | 0 | 1
  HPV-59 M24: number analyzed (Participants) | 1298 | 1246
  HPV-59 M24 | 1 | 1
  HPV-66 M24: number analyzed (Participants) | 1289 | 1238
  HPV-66 M24 | 0 | 1
  HPV-68 M24: number analyzed (Participants) | 1281 | 1240
  HPV-68 M24 | 2 | 0
  HPV-31/33/45 M24: number analyzed (Participants) | 1305 | 1261
  HPV-31/33/45 M24 | 3 | 1
  HPV-16/18/31/33/45 M24: number analyzed (Participants) | 1305 | 1262
  HPV-16/18/31/33/45 M24 | 3 | 3
  HRW-HPV M24: number analyzed (Participants) | 1305 | 1262
  HRW-HPV M24 | 21 | 14
  HR-HPV M24: number analyzed (Participants) | 1305 | 1262
  HR-HPV M24 | 21 | 15
  HPV-16 M48: number analyzed (Participants) | 2575 | 2587
  HPV-16 M48 | 1 | 17
  HPV-18 M48: number analyzed (Participants) | 2633 | 2639
  HPV-18 M48 | 0 | 5
  HPV-31 M48: number analyzed (Participants) | 2640 | 2643
  HPV-31 M48 | 3 | 11
  HPV-33 M48: number analyzed (Participants) | 2632 | 2643
  HPV-33 M48 | 6 | 6
  HPV-35 M48: number analyzed (Participants) | 2655 | 2662
  HPV-35 M48 | 5 | 7
  HPV-39 M48: number analyzed (Participants) | 2611 | 2632
  HPV-39 M48 | 12 | 16
  HPV-45 M48: number analyzed (Participants) | 2643 | 2661
  HPV-45 M48 | 4 | 1
  HPV-51 M48: number analyzed (Participants) | 2610 | 2615
  HPV-51 M48 | 20 | 16
  HPV-52 M48: number analyzed (Participants) | 2527 | 2538
  HPV-52 M48 | 41 | 40
  HPV-56 M48: number analyzed (Participants) | 2635 | 2639
  HPV-56 M48 | 11 | 5
  HPV-58 M48: number analyzed (Participants) | 2626 | 2629
  HPV-58 M48 | 4 | 9
  HPV-59 M48: number analyzed (Participants) | 2663 | 2654
  HPV-59 M48 | 5 | 2
  HPV-66 M48: number analyzed (Participants) | 2633 | 2624
  HPV-66 M48 | 8 | 7
  HPV-68 M48: number analyzed (Participants) | 2629 | 2643
  HPV-68 M48 | 9 | 4
  HPV-31/33/45 M48: number analyzed (Participants) | 2672 | 2680
  HPV-31/33/45 M48 | 12 | 18
  HPV-16/18/31/33/45 M48: number analyzed (Participants) | 2672 | 2681
  HPV-16/18/31/33/45 M48 | 13 | 40
  HRW-HPV M48: number analyzed (Participants) | 2672 | 2681
  HRW-HPV M48 | 122 | 119
  HR-HPV M48: number analyzed (Participants) | 2672 | 2681
  HR-HPV M48 | 122 | 137
  HPV-16 M57: number analyzed (Participants) | 2604 | 2620
  HPV-16 M57 | 1 | 29
  HPV-18 M57: number analyzed (Participants) | 2664 | 2672
  HPV-18 M57 | 0 | 8
  HPV-31 M57: number analyzed (Participants) | 2671 | 2676
  HPV-31 M57 | 3 | 16
  HPV-33 M57: number analyzed (Participants) | 2663 | 2675
  HPV-33 M57 | 8 | 9
  HPV-35 M57: number analyzed (Participants) | 2686 | 2695
  HPV-35 M57 | 11 | 9
  HPV-39 M57: number analyzed (Participants) | 2641 | 2664
  HPV-39 M57 | 25 | 22
  HPV-45 M57: number analyzed (Participants) | 2674 | 2694
  HPV-45 M57 | 5 | 2
  HPV-51 M57: number analyzed (Participants) | 2639 | 2647
  HPV-51 M57 | 28 | 24
  HPV-52 M57: number analyzed (Participants) | 2553 | 2569
  HPV-52 M57 | 70 | 63
  HPV-56 M57: number analyzed (Participants) | 2665 | 2672
  HPV-56 M57 | 14 | 11
  HPV-58 M57: number analyzed (Participants) | 2656 | 2661
  HPV-58 M57 | 15 | 18
  HPV-59 M57: number analyzed (Participants) | 2694 | 2687
  HPV-59 M57 | 7 | 2
  HPV-66 M57: number analyzed (Participants) | 2662 | 2657
  HPV-66 M57 | 17 | 10
  HPV-68 M57: number analyzed (Participants) | 2659 | 2675
  HPV-68 M57 | 12 | 12
  HPV-31/33/45 M57: number analyzed (Participants) | 2703 | 2713
  HPV-31/33/45 M57 | 15 | 27
  HPV-16/18/31/33/45 M57 | 16 | 63
  HRW-HPV M57 | 192 | 188
  HR-HPV M57 | 192 | 215
  HPV-16 M72: number analyzed (Participants) | 2607 | 2622
  HPV-16 M72 | 1 | 30
  HPV-18 M72: number analyzed (Participants) | 2666 | 2675
  HPV-18 M72 | 0 | 8
  HPV-31 M72: number analyzed (Participants) | 2674 | 2679
  HPV-31 M72 | 3 | 16
  HPV-33 M72: number analyzed (Participants) | 2666 | 2678
  HPV-33 M72 | 9 | 9
  HPV-35 M72: number analyzed (Participants) | 2689 | 2698
  HPV-35 M72 | 12 | 9
  HPV-39 M72: number analyzed (Participants) | 2643 | 2667
  HPV-39 M72 | 25 | 22
  HPV-45 M72: number analyzed (Participants) | 2677 | 2697
  HPV-45 M72 | 5 | 2
  HPV-51 M72: number analyzed (Participants) | 2642 | 2650
  HPV-51 M72 | 28 | 25
  HPV-52 M72: number analyzed (Participants) | 2555 | 2571
  HPV-52 M72 | 72 | 65
  HPV-56 M72: number analyzed (Participants) | 2667 | 2675
  HPV-56 M72 | 14 | 12
  HPV-58 M72: number analyzed (Participants) | 2659 | 2664
  HPV-58 M72 | 15 | 18
  HPV-59 M72: number analyzed (Participants) | 2697 | 2690
  HPV-59 M72 | 8 | 2
  HPV-66 M72: number analyzed (Participants) | 2665 | 2660
  HPV-66 M72 | 17 | 10
  HPV-68 M72: number analyzed (Participants) | 2662 | 2678
  HPV-68 M72 | 12 | 12
  HPV-31/33/45 M72: number analyzed (Participants) | 2706 | 2716
  HPV-31/33/45 M72 | 16 | 27
  HPV-16/18/31/33/45 M72 | 17 | 64
  HRW-HPV M72 | 196 | 192
  HR-HPV M72 | 196 | 219

11. Secondary Outcome: Number of Subjects With Any Cytological Abnormality Including Atypical Squamous Cells of Undetermined Significance (ASC-US+) Associated With HPV-16 and/or HPV-18 Cervical Infection
Description: Cytological abnormalities = atypical squamous cells of undetermined significance (ASC-DNA- and sero-: subjects HPV DNA negative at Months 0 and 6 by PCR and seronegative at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA) Overall: subjects DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus. US).
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2803 | 2802
Participants
  Sero negative, DNA negative HPV-16/18 M24: number analyzed (Participants) | 2494 | 2502
  Sero negative, DNA negative HPV-16/18 M24 | 1 | 16
  Sero negative, DNA negative HPV-16 M24: number analyzed (Participants) | 1935 | 1884
  Sero negative, DNA negative HPV-16 M24 | 1 | 12
  Sero negative, DNA negative HPV-18 M24: number analyzed (Participants) | 2318 | 2314
  Sero negative, DNA negative HPV-18 M24 | 0 | 5
  Overall, HPV-16/18 M24: number analyzed (Participants) | 2772 | 2763
  Overall, HPV-16/18 M24 | 3 | 24
  Overall, HPV-16 M24: number analyzed (Participants) | 2674 | 2671
  Overall, HPV-16 M24 | 3 | 17
  Overall, HPV-18 M24: number analyzed (Participants) | 2736 | 2730
  Overall, HPV-18 M24 | 0 | 8
  Sero negative, DNA negative HPV-16/18 M48: number analyzed (Participants) | 2520 | 2531
  Sero negative, DNA negative HPV-16/18 M48 | 2 | 39
  Sero negative, DNA negative HPV-16 M48: number analyzed (Participants) | 1957 | 1908
  Sero negative, DNA negative HPV-16 M48 | 2 | 28
  Sero negative, DNA negative HPV-18 M48: number analyzed (Participants) | 2342 | 2340
  Sero negative, DNA negative HPV-18 M48 | 0 | 12
  Overall, HPV-16/18 M48: number analyzed (Participants) | 2801 | 2799
  Overall, HPV-16/18 M48 | 5 | 53
  Overall, HPV-16 M48: number analyzed (Participants) | 2703 | 2707
  Overall, HPV-16 M48 | 4 | 39
  Overall, HPV-18 M48: number analyzed (Participants) | 2764 | 2765
  Overall, HPV-18 M48 | 1 | 16
  Sero negative, DNA negative HPV-16/18 M57: number analyzed (Participants) | 2522 | 2535
  Sero negative, DNA negative HPV-16/18 M57 | 4 | 53
  Sero negative, DNA negative HPV-16 M57: number analyzed (Participants) | 1958 | 1909
  Sero negative, DNA negative HPV-16 M57 | 3 | 38
  Sero negative, DNA negative HPV-18 M57: number analyzed (Participants) | 2344 | 2344
  Sero negative, DNA negative HPV-18 M57 | 1 | 16
  Overall, HPV-16/18 M57 | 10 | 71
  Overall, HPV-16 M57: number analyzed (Participants) | 2705 | 2710
  Overall, HPV-16 M57 | 7 | 52
  Overall, HPV-18 M57: number analyzed (Participants) | 2766 | 2768
  Overall, HPV-18 M57 | 3 | 21
  Sero negative, DNA negative HPV-16/18 M72: number analyzed (Participants) | 2521 | 2534
  Sero negative, DNA negative HPV-16/18 M72 | 5 | 60
  Sero negative, DNA negative HPV-16 M72: number analyzed (Participants) | 1957 | 1908
  Sero negative, DNA negative HPV-16 M72 | 4 | 44
  Sero negative, DNA negative HPV-18 M72: number analyzed (Participants) | 2343 | 2344
  Sero negative, DNA negative HPV-18 M72 | 1 | 17
  Overall, HPV-16/18 M72: number analyzed (Participants) | 2802 | 2801
  Overall, HPV-16/18 M72 | 12 | 83
  Overall, HPV-16 M72: number analyzed (Participants) | 2704 | 2709
  Overall, HPV-16 M72 | 9 | 62
  Overall, HPV-18 M72: number analyzed (Participants) | 2765 | 2767
  Overall, HPV-18 M72 | 3 | 24

12. Secondary Outcome: Number of Subjects With Any Cytological Abnormality Including Atypical Squamous Cells of Undetermined Significance (ASC-US+) Associated With Any Oncogenic HPV Type
Description: Cytological abnormalities = atypical squamous cells of undetermined significance (ASC-US). Oncogenic HPV types assessed were HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68 individually or in combination. Subjects were HPV DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus. HRW-HPV=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HR-HPV=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2808 | 2812
Participants
  HPV-16 M24: number analyzed (Participants) | 2674 | 2671
  HPV-16 M24 | 3 | 17
  HPV-18 M24: number analyzed (Participants) | 2736 | 2730
  HPV-18 M24 | 0 | 8
  HPV-31 M24: number analyzed (Participants) | 2741 | 2732
  HPV-31 M24 | 5 | 7
  HPV-33 M24: number analyzed (Participants) | 2734 | 2732
  HPV-33 M24 | 5 | 7
  HPV-35 M24: number analyzed (Participants) | 2760 | 2752
  HPV-35 M24 | 6 | 4
  HPV-39 M24: number analyzed (Participants) | 2712 | 2722
  HPV-39 M24 | 11 | 8
  HPV-45 M24: number analyzed (Participants) | 2747 | 2750
  HPV-45 M24 | 4 | 5
  HPV-51 M24: number analyzed (Participants) | 2709 | 2707
  HPV-51 M24 | 19 | 17
  HPV-52 M24: number analyzed (Participants) | 2622 | 2614
  HPV-52 M24 | 29 | 16
  HPV-56 M24: number analyzed (Participants) | 2737 | 2730
  HPV-56 M24 | 9 | 13
  HPV-58 M24: number analyzed (Participants) | 2726 | 2717
  HPV-58 M24 | 9 | 11
  HPV-59 M24: number analyzed (Participants) | 2767 | 2745
  HPV-59 M24 | 8 | 4
  HPV-66 M24: number analyzed (Participants) | 2733 | 2714
  HPV-66 M24 | 12 | 9
  HPV-68 M24: number analyzed (Participants) | 2728 | 2733
  HPV-68 M24 | 10 | 10
  HPV-31/33/45 M24: number analyzed (Participants) | 2776 | 2772
  HPV-31/33/45 M24 | 13 | 18
  HPV-16/18/31/33/45 M24: number analyzed (Participants) | 2776 | 2773
  HPV-16/18/31/33/45 M24 | 15 | 42
  HRW-HPV M24: number analyzed (Participants) | 2776 | 2773
  HRW-HPV M24 | 88 | 90
  HR-HPV M24: number analyzed (Participants) | 2776 | 2773
  HR-HPV M24 | 90 | 105
  HPV-16 M48: number analyzed (Participants) | 2703 | 2707
  HPV-16 M48 | 4 | 39
  HPV-18 M48: number analyzed (Participants) | 2764 | 2765
  HPV-18 M48 | 1 | 16
  HPV-31 M48: number analyzed (Participants) | 2770 | 2767
  HPV-31 M48 | 10 | 21
  HPV-33 M48: number analyzed (Participants) | 2763 | 2768
  HPV-33 M48 | 11 | 20
  HPV-35 M48: number analyzed (Participants) | 2789 | 2788
  HPV-35 M48 | 12 | 15
  HPV-39 M48: number analyzed (Participants) | 2742 | 2757
  HPV-39 M48 | 29 | 21
  HPV-45 M48: number analyzed (Participants) | 2777 | 2786
  HPV-45 M48 | 6 | 6
  HPV-51 M48: number analyzed (Participants) | 2737 | 2741
  HPV-51 M48 | 42 | 47
  HPV-52 M48: number analyzed (Participants) | 2650 | 2649
  HPV-52 M48 | 54 | 45
  HPV-56 M48: number analyzed (Participants) | 2766 | 2765
  HPV-56 M48 | 25 | 27
  HPV-58 M48: number analyzed (Participants) | 2755 | 2753
  HPV-58 M48 | 20 | 20
  HPV-59 M48: number analyzed (Participants) | 2797 | 2781
  HPV-59 M48 | 17 | 10
  HPV-66 M48: number analyzed (Participants) | 2763 | 2750
  HPV-66 M48 | 27 | 20
  HPV-68 M48: number analyzed (Participants) | 2758 | 2769
  HPV-68 M48 | 22 | 19
  HPV-31/33/45 M48: number analyzed (Participants) | 2806 | 2808
  HPV-31/33/45 M48 | 24 | 41
  HPV-16/18/31/33/45 M48: number analyzed (Participants) | 2806 | 2809
  HPV-16/18/31/33/45 M48 | 28 | 92
  HRW-HPV M48: number analyzed (Participants) | 2806 | 2809
  HRW-HPV M48 | 196 | 212
  HR-HPV M48: number analyzed (Participants) | 2806 | 2809
  HR-HPV M48 | 199 | 238
  HPV-16 M57: number analyzed (Participants) | 2705 | 2710
  HPV-16 M57 | 7 | 52
  HPV-18 M57: number analyzed (Participants) | 2766 | 2768
  HPV-18 M57 | 3 | 21
  HPV-31 M57: number analyzed (Participants) | 2772 | 2770
  HPV-31 M57 | 12 | 28
  HPV-33 M57: number analyzed (Participants) | 2765 | 2771
  HPV-33 M57 | 15 | 29
  HPV-35 M57: number analyzed (Participants) | 2791 | 2791
  HPV-35 M57 | 18 | 19
  HPV-39 M57: number analyzed (Participants) | 2744 | 2760
  HPV-39 M57 | 40 | 31
  HPV-45 M57: number analyzed (Participants) | 2779 | 2789
  HPV-45 M57 | 9 | 12
  HPV-51 M57: number analyzed (Participants) | 2739 | 2743
  HPV-51 M57 | 57 | 64
  HPV-52 M57: number analyzed (Participants) | 2652 | 2652
  HPV-52 M57 | 71 | 74
  HPV-56 M57: number analyzed (Participants) | 2768 | 2767
  HPV-56 M57 | 39 | 43
  HPV-58 M57: number analyzed (Participants) | 2757 | 2756
  HPV-58 M57 | 34 | 42
  HPV-59 M57: number analyzed (Participants) | 2799 | 2784
  HPV-59 M57 | 19 | 15
  HPV-66 M57: number analyzed (Participants) | 2765 | 2752
  HPV-66 M57 | 39 | 39
  HPV-68 M57: number analyzed (Participants) | 2760 | 2772
  HPV-68 M57 | 28 | 30
  HPV-31/33/45 M57: number analyzed (Participants) | 2808 | 2811
  HPV-31/33/45 M57 | 32 | 61
  HPV-16/18/31/33/45 M57 | 41 | 127
  HRW-HPV M57 | 127 | 274
  HR-HPV M57 | 278 | 343
  HPV-16 M72: number analyzed (Participants) | 2704 | 2709
  HPV-16 M72 | 9 | 62
  HPV-18 M72: number analyzed (Participants) | 2765 | 2767
  HPV-18 M72 | 3 | 25
  HPV-31 M72: number analyzed (Participants) | 2771 | 2769
  HPV-31 M72 | 12 | 32
  HPV-33 M72: number analyzed (Participants) | 2764 | 2770
  HPV-33 M72 | 17 | 32
  HPV-35 M72: number analyzed (Participants) | 2790 | 2790
  HPV-35 M72 | 20 | 21
  HPV-39 M72: number analyzed (Participants) | 2743 | 2759
  HPV-39 M72 | 49 | 35
  HPV-45 M72: number analyzed (Participants) | 2778 | 2788
  HPV-45 M72 | 9 | 12
  HPV-51 M72: number analyzed (Participants) | 2738 | 2742
  HPV-51 M72 | 64 | 78
  HPV-52 M72: number analyzed (Participants) | 2651 | 2651
  HPV-52 M72 | 83 | 81
  HPV-56 M72: number analyzed (Participants) | 2767 | 2766
  HPV-56 M72 | 46 | 51
  HPV-58 M72: number analyzed (Participants) | 2756 | 2756
  HPV-58 M72 | 36 | 49
  HPV-59 M72: number analyzed (Participants) | 2798 | 2783
  HPV-59 M72 | 20 | 17
  HPV-66 M72: number analyzed (Participants) | 2764 | 2751
  HPV-66 M72 | 42 | 46
  HPV-68 M72: number analyzed (Participants) | 2759 | 2771
  HPV-68 M72 | 30 | 37
  HPV-31/33/45 M72: number analyzed (Participants) | 2807 | 2810
  HPV-31/33/45 M72 | 34 | 66
  HPV-16/18/31/33/45 M72: number analyzed (Participants) | 2807 | 2811
  HPV-16/18/31/33/45 M72 | 45 | 144
  HRW-HPV M72: number analyzed (Participants) | 2807 | 2811
  HRW-HPV M72 | 309 | 352
  HR-HPV M72: number analyzed (Participants) | 2807 | 2811
  HR-HPV M72 | 313 | 386

13. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN1+ Associated With HPV-16 and/or HPV-18 Cervical Infection
Description: CIN1+ = CIN grades 1, 2, and3, low-grade cervical glandular intraepithelial neoplasia (LCGIN), high grade cervical glandular intraepithelial neoplasia (HCGIN), adenocarcinoma in-situ (AIS) or invasive cervical cancer. DNA- and sero-: subjects HPV DNA negative at Months 0 and 6 by PCR and seronegative at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA) Overall: subjects DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2805 | 2802
Participants
  Sero negative, DNA negative HPV-16/18 M24: number analyzed (Participants) | 2497 | 2502
  Sero negative, DNA negative HPV-16/18 M24 | 0 | 4
  Sero negative, DNA negative HPV-16 M24: number analyzed (Participants) | 1937 | 1884
  Sero negative, DNA negative HPV-16 M24 | 0 | 4
  Sero negative, DNA negative HPV-18 M24: number analyzed (Participants) | 2320 | 2314
  Sero negative, DNA negative HPV-18 M24 | 0 | 0
  Overall, HPV-16/18 M24: number analyzed (Participants) | 2775 | 2764
  Overall, HPV-16/18 M24 | 0 | 5
  Overall, HPV-16 M24: number analyzed (Participants) | 2677 | 2672
  Overall, HPV-16 M24 | 0 | 5
  Overall, HPV-18 M24: number analyzed (Participants) | 2738 | 2731
  Overall, HPV-18 M24 | 0 | 0
  Sero negative, DNA negative HPV-16/18 M48: number analyzed (Participants) | 2522 | 2531
  Sero negative, DNA negative HPV-16/18 M48 | 1 | 12
  Sero negative, DNA negative HPV-16 M48: number analyzed (Participants) | 1958 | 1908
  Sero negative, DNA negative HPV-16 M48 | 1 | 8
  Sero negative, DNA negative HPV-18 M48: number analyzed (Participants) | 2344 | 2340
  Sero negative, DNA negative HPV-18 M48 | 0 | 4
  Overall, HPV-16/18 M48: number analyzed (Participants) | 2803 | 2799
  Overall, HPV-16/18 M48 | 1 | 14
  Overall, HPV-16 M48: number analyzed (Participants) | 2705 | 2707
  Overall, HPV-16 M48 | 1 | 10
  Overall, HPV-18 M48: number analyzed (Participants) | 2766 | 2765
  Overall, HPV-18 M48 | 0 | 4
  Sero negative, DNA negative HPV-16/18 M57: number analyzed (Participants) | 2524 | 2535
  Sero negative, DNA negative HPV-16/18 M57 | 1 | 15
  Sero negative, DNA negative HPV-16 M57: number analyzed (Participants) | 1959 | 1909
  Sero negative, DNA negative HPV-16 M57 | 1 | 10
  Sero negative, DNA negative HPV-18 M57: number analyzed (Participants) | 2346 | 2344
  Sero negative, DNA negative HPV-18 M57 | 0 | 5
  Overall, HPV-16/18 M57 | 1 | 18
  Overall, HPV-16 M57: number analyzed (Participants) | 2707 | 2710
  Overall, HPV-16 M57 | 1 | 13
  Overall, HPV-18 M57: number analyzed (Participants) | 2768 | 2768
  Overall, HPV-18 M57 | 0 | 5
  Sero negative, DNA negative HPV-16/18 M72: number analyzed (Participants) | 2523 | 2534
  Sero negative, DNA negative HPV-16/18 M72 | 1 | 15
  Sero negative, DNA negative HPV-16 M72: number analyzed (Participants) | 1958 | 1908
  Sero negative, DNA negative HPV-16 M72 | 1 | 10
  Sero negative, DNA negative HPV-18 M72: number analyzed (Participants) | 2345 | 2344
  Sero negative, DNA negative HPV-18 M72 | 0 | 5
  Overall, HPV-16/18 M72: number analyzed (Participants) | 2804 | 2801
  Overall, HPV-16/18 M72 | 1 | 18
  Overall, HPV-16 M72: number analyzed (Participants) | 2706 | 2709
  Overall, HPV-16 M72 | 1 | 13
  Overall, HPV-18 M72: number analyzed (Participants) | 2767 | 2767
  Overall, HPV-18 M72 | 0 | 5

14. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN2+ Associated With HPV-16 and/or HPV-18 Cervical Infection
Description: CIN2+ = CIN grades 2 and 3, LCGIN, HCGIN, AIS or invasive cervical cancer. DNA- and sero-: subjects HPV DNA negative at Months 0 and 6 by PCR and seronegative at Month 0 for the corresponding HPV-type by Enzyme-linked Immunosorbent Assay (ELISA) Overall: subjects DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2805 | 2802
Participants
  Sero negative, DNA negative HPV-16/18 M24: number analyzed (Participants) | 2497 | 2502
  Sero negative, DNA negative HPV-16/18 M24 | 0 | 3
  Sero negative, DNA negative HPV-16 M24: number analyzed (Participants) | 1937 | 1884
  Sero negative, DNA negative HPV-16 M24 | 0 | 3
  Sero negative, DNA negative HPV-18 M24: number analyzed (Participants) | 2320 | 2314
  Sero negative, DNA negative HPV-18 M24 | 0 | 0
  Overall, HPV-16/18 M24: number analyzed (Participants) | 2775 | 2764
  Overall, HPV-16/18 M24 | 0 | 4
  Overall, HPV-16 M24: number analyzed (Participants) | 2677 | 2672
  Overall, HPV-16 M24 | 0 | 4
  Overall, HPV-18 M24: number analyzed (Participants) | 2738 | 2731
  Overall, HPV-18 M24 | 0 | 0
  Sero negative, DNA negative HPV-16/18 M48: number analyzed (Participants) | 2522 | 2531
  Sero negative, DNA negative HPV-16/18 M48 | 1 | 6
  Sero negative, DNA negative HPV-16 M48: number analyzed (Participants) | 1958 | 1908
  Sero negative, DNA negative HPV-16 M48 | 1 | 6
  Sero negative, DNA negative HPV-18 M48: number analyzed (Participants) | 2344 | 2340
  Sero negative, DNA negative HPV-18 M48 | 0 | 0
  Overall, HPV-16/18 M48: number analyzed (Participants) | 2803 | 2799
  Overall, HPV-16/18 M48 | 1 | 7
  Overall, HPV-16 M48: number analyzed (Participants) | 2705 | 2707
  Overall, HPV-16 M48 | 1 | 7
  Overall, HPV-18 M48: number analyzed (Participants) | 2766 | 2765
  Overall, HPV-18 M48 | 0 | 0
  Sero negative, DNA negative HPV-16/18 M57: number analyzed (Participants) | 2524 | 2535
  Sero negative, DNA negative HPV-16/18 M57 | 1 | 8
  Sero negative, DNA negative HPV-16 M57: number analyzed (Participants) | 1959 | 1909
  Sero negative, DNA negative HPV-16 M57 | 1 | 8
  Sero negative, DNA negative HPV-18 M57: number analyzed (Participants) | 2346 | 2344
  Sero negative, DNA negative HPV-18 M57 | 0 | 0
  Overall, HPV-16/18 M57 | 1 | 10
  Overall, HPV-16 M57: number analyzed (Participants) | 2707 | 2710
  Overall, HPV-16 M57 | 1 | 10
  Overall, HPV-18 M57: number analyzed (Participants) | 2768 | 2768
  Overall, HPV-18 M57 | 0 | 0
  Sero negative, DNA negative HPV-16/18 M72: number analyzed (Participants) | 2523 | 2534
  Sero negative, DNA negative HPV-16/18 M72 | 1 | 8
  Sero negative, DNA negative HPV-16 M72: number analyzed (Participants) | 1958 | 1908
  Sero negative, DNA negative HPV-16 M72 | 1 | 8
  Sero negative, DNA negative HPV-18 M72: number analyzed (Participants) | 2345 | 2344
  Sero negative, DNA negative HPV-18 M72 | 0 | 0
  Overall, HPV-16/18 M72: number analyzed (Participants) | 2804 | 2801
  Overall, HPV-16/18 M72 | 1 | 10
  Overall, HPV-16 M72: number analyzed (Participants) | 2706 | 2709
  Overall, HPV-16 M72 | 1 | 10
  Overall, HPV-18 M72: number analyzed (Participants) | 2767 | 2767
  Overall, HPV-18 M72 | 0 | 0

15. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN1+ Associated With Cervical Infection With Any Oncogenic HPV Type
Description: CIN1+ = CIN grades 1, 2 and 3, LCGIN, HCGIN, AIS or invasive cervical cancer. Oncogenic HPV types assessed were HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68 individually or in combination. Subjects were HPV DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus. HRW-HPV=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HR-HPV=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2810 | 2812
Participants
  HPV-16 M24: number analyzed (Participants) | 2677 | 2672
  HPV-16 M24 | 0 | 5
  HPV-18 M24: number analyzed (Participants) | 2738 | 2731
  HPV-18 M24 | 0 | 0
  HPV-31 M24: number analyzed (Participants) | 2744 | 2733
  HPV-31 M24 | 0 | 1
  HPV-33 M24: number analyzed (Participants) | 2737 | 2733
  HPV-33 M24 | 2 | 1
  HPV-35 M24: number analyzed (Participants) | 2763 | 2753
  HPV-35 M24 | 1 | 1
  HPV-39 M24: number analyzed (Participants) | 2714 | 2723
  HPV-39 M24 | 2 | 0
  HPV-45 M24: number analyzed (Participants) | 2750 | 2751
  HPV-45 M24 | 2 | 1
  HPV-51 M24: number analyzed (Participants) | 2711 | 2708
  HPV-51 M24 | 1 | 3
  HPV-52 M24: number analyzed (Participants) | 2624 | 2615
  HPV-52 M24 | 2 | 3
  HPV-56 M24: number analyzed (Participants) | 2739 | 2731
  HPV-56 M24 | 0 | 2
  HPV-58 M24: number analyzed (Participants) | 2729 | 2718
  HPV-58 M24 | 0 | 1
  HPV-59 M24: number analyzed (Participants) | 2770 | 2746
  HPV-59 M24 | 1 | 0
  HPV-66 M24: number analyzed (Participants) | 2736 | 2715
  HPV-66 M24 | 3 | 2
  HPV-68 M24: number analyzed (Participants) | 2731 | 2734
  HPV-68 M24 | 0 | 2
  HPV-31/33/45 M24: number analyzed (Participants) | 2779 | 2773
  HPV-31/33/45 M24 | 3 | 3
  HPV-16/18/31/33/45 M24: number analyzed (Participants) | 2779 | 2774
  HPV-16/18/31/33/45 M24 | 3 | 8
  HRW-HPV M24: number analyzed (Participants) | 2779 | 2774
  HRW-HPV M24 | 11 | 14
  HR-HPV M24: number analyzed (Participants) | 2779 | 2774
  HR-HPV M24 | 11 | 17
  HPV-16 M48: number analyzed (Participants) | 2705 | 2707
  HPV-16 M48 | 1 | 10
  HPV-18 M48: number analyzed (Participants) | 2766 | 2765
  HPV-18 M48 | 0 | 4
  HPV-31 M48: number analyzed (Participants) | 2772 | 2767
  HPV-31 M48 | 0 | 4
  HPV-33 M48: number analyzed (Participants) | 2765 | 2768
  HPV-33 M48 | 3 | 2
  HPV-35 M48: number analyzed (Participants) | 2791 | 2788
  HPV-35 M48 | 1 | 3
  HPV-39 M48: number analyzed (Participants) | 2743 | 2757
  HPV-39 M48 | 4 | 1
  HPV-45 M48: number analyzed (Participants) | 2779 | 2786
  HPV-45 M48 | 3 | 1
  HPV-51 M48: number analyzed (Participants) | 2739 | 2741
  HPV-51 M48 | 1 | 8
  HPV-52 M48: number analyzed (Participants) | 2651 | 2649
  HPV-52 M48 | 7 | 9
  HPV-56 M48: number analyzed (Participants) | 2768 | 2765
  HPV-56 M48 | 1 | 3
  HPV-58 M48: number analyzed (Participants) | 2757 | 2753
  HPV-58 M48 | 4 | 4
  HPV-59 M48: number analyzed (Participants) | 2799 | 2781
  HPV-59 M48 | 1 | 0
  HPV-66 M48: number analyzed (Participants) | 2765 | 2750
  HPV-66 M48 | 6 | 3
  HPV-68 M48: number analyzed (Participants) | 2760 | 2769
  HPV-68 M48 | 2 | 2
  HPV-31/33/45 M48: number analyzed (Participants) | 2808 | 2808
  HPV-31/33/45 M48 | 5 | 7
  HPV-16/18/31/33/45 M48: number analyzed (Participants) | 2808 | 2809
  HPV-16/18/31/33/45 M48 | 6 | 21
  HRW-HPV M48: number analyzed (Participants) | 2808 | 2809
  HRW-HPV M48 | 27 | 35
  HR-HPV M48: number analyzed (Participants) | 2808 | 2809
  HR-HPV M48 | 27 | 44
  HPV-16 M57: number analyzed (Participants) | 2707 | 2710
  HPV-16 M57 | 1 | 13
  HPV-18 M57: number analyzed (Participants) | 2768 | 2768
  HPV-18 M57 | 0 | 5
  HPV-31 M57: number analyzed (Participants) | 2774 | 2770
  HPV-31 M57 | 0 | 6
  HPV-33 M57: number analyzed (Participants) | 2767 | 2771
  HPV-33 M57 | 3 | 2
  HPV-35 M57: number analyzed (Participants) | 2793 | 2791
  HPV-35 M57 | 2 | 3
  HPV-39 M57: number analyzed (Participants) | 2745 | 2760
  HPV-39 M57 | 7 | 1
  HPV-45 M57: number analyzed (Participants) | 2781 | 2789
  HPV-45 M57 | 3 | 3
  HPV-51 M57: number analyzed (Participants) | 2741 | 2743
  HPV-51 M57 | 2 | 9
  HPV-52 M57: number analyzed (Participants) | 2653 | 2652
  HPV-52 M57 | 11 | 11
  HPV-56 M57: number analyzed (Participants) | 2770 | 2767
  HPV-56 M57 | 2 | 4
  HPV-58 M57: number analyzed (Participants) | 2759 | 2756
  HPV-58 M57 | 4 | 9
  HPV-59 M57: number analyzed (Participants) | 2801 | 2784
  HPV-59 M57 | 1 | 0
  HPV-66 M57: number analyzed (Participants) | 2767 | 2752
  HPV-66 M57 | 6 | 5
  HPV-68 M57: number analyzed (Participants) | 2762 | 2772
  HPV-68 M57 | 3 | 3
  HPV-31/33/45 M57: number analyzed (Participants) | 2810 | 2811
  HPV-31/33/45 M57 | 5 | 10
  HPV-16/18/31/33/45 M57 | 6 | 27
  HRW-HPV M57 | 37 | 49
  HR-HPV M57 | 37 | 60
  HPV-16 M72: number analyzed (Participants) | 2706 | 2709
  HPV-16 M72 | 1 | 13
  HPV-18 M72: number analyzed (Participants) | 2767 | 2767
  HPV-18 M72 | 0 | 5
  HPV-31 M72: number analyzed (Participants) | 2773 | 2769
  HPV-31 M72 | 0 | 6
  HPV-33 M72: number analyzed (Participants) | 2766 | 2770
  HPV-33 M72 | 5 | 3
  HPV-35 M72: number analyzed (Participants) | 2792 | 2790
  HPV-35 M72 | 2 | 3
  HPV-39 M72: number analyzed (Participants) | 2744 | 2759
  HPV-39 M72 | 7 | 1
  HPV-45 M72: number analyzed (Participants) | 2780 | 2788
  HPV-45 M72 | 3 | 3
  HPV-51 M72: number analyzed (Participants) | 2740 | 2742
  HPV-51 M72 | 3 | 9
  HPV-52 M72: number analyzed (Participants) | 2652 | 2651
  HPV-52 M72 | 11 | 12
  HPV-56 M72: number analyzed (Participants) | 2769 | 2766
  HPV-56 M72 | 2 | 4
  HPV-58 M72: number analyzed (Participants) | 2758 | 2755
  HPV-58 M72 | 6 | 9
  HPV-59 M72: number analyzed (Participants) | 2800 | 2783
  HPV-59 M72 | 1 | 0
  HPV-66 M72: number analyzed (Participants) | 2766 | 2751
  HPV-66 M72 | 6 | 8
  HPV-68 M72: number analyzed (Participants) | 2761 | 2771
  HPV-68 M72 | 3 | 3
  HPV-31/33/45 M72: number analyzed (Participants) | 2809 | 2810
  HPV-31/33/45 M72 | 7 | 11
  HPV-16/18/31/33/45 M72: number analyzed (Participants) | 2809 | 2811
  HPV-16/18/31/33/45 M72 | 8 | 28
  HRW-HPV M72: number analyzed (Participants) | 2809 | 2811
  HRW-HPV M72 | 42 | 53
  HR-HPV M72: number analyzed (Participants) | 2809 | 2811
  HR-HPV M72 | 42 | 64

16. Secondary Outcome: Number of Subjects With Histopathologically-confirmed CIN2+ Associated With Cervical Infection With Any Oncogenic HPV Type
Description: CIN2+ = CIN grades 2 and 3, LCGIN, HCGIN, AIS or invasive cervical cancer. Oncogenic HPV types assessed were HPV-16, -18, -31, -33, -35, -39, -45, -51, -52, -56, -58, -59, -66 and -68 individually or in combination. Subjects were HPV DNA- at Months 0 and 6 for the corresponding HPV-type, regardless of initial serostatus. HRW-HPV=All high-risk (oncogenic) HPV types excluding HPV-16 and HPV-18 HR-HPV=High-risk (oncogenic) HPV types: HPV-16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59, 66 and 68.
Time Frame: At Months 24, 48, 57 and 72
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 2810 | 2812
Participants
  HPV-16 M24: number analyzed (Participants) | 2677 | 2672
  HPV-16 M24 | 0 | 4
  HPV-18 M24: number analyzed (Participants) | 2738 | 2731
  HPV-18 M24 | 0 | 0
  HPV-31 M24: number analyzed (Participants) | 2744 | 2733
  HPV-31 M24 | 0 | 0
  HPV-33 M24: number analyzed (Participants) | 2737 | 2733
  HPV-33 M24 | 1 | 1
  HPV-35 M24: number analyzed (Participants) | 2763 | 2753
  HPV-35 M24 | 0 | 0
  HPV-39 M24: number analyzed (Participants) | 2714 | 2723
  HPV-39 M24 | 0 | 0
  HPV-45 M24: number analyzed (Participants) | 2750 | 2751
  HPV-45 M24 | 0 | 0
  HPV-51 M24: number analyzed (Participants) | 2711 | 2708
  HPV-51 M24 | 0 | 0
  HPV-52 M24: number analyzed (Participants) | 2624 | 2615
  HPV-52 M24 | 0 | 0
  HPV-56 M24: number analyzed (Participants) | 2739 | 2731
  HPV-56 M24 | 0 | 0
  HPV-58 M24: number analyzed (Participants) | 2729 | 2718
  HPV-58 M24 | 0 | 1
  HPV-59 M24: number analyzed (Participants) | 2770 | 2746
  HPV-59 M24 | 0 | 0
  HPV-66 M24: number analyzed (Participants) | 2736 | 2715
  HPV-66 M24 | 1 | 1
  HPV-68 M24: number analyzed (Participants) | 2731 | 2734
  HPV-68 M24 | 0 | 0
  HPV-31/33/45 M24: number analyzed (Participants) | 2779 | 2773
  HPV-31/33/45 M24 | 1 | 1
  HPV-16/18/31/33/45 M24: number analyzed (Participants) | 2779 | 2774
  HPV-16/18/31/33/45 M24 | 1 | 5
  HRW-HPV M24: number analyzed (Participants) | 2779 | 2774
  HRW-HPV M24 | 2 | 3
  HR-HPV M24: number analyzed (Participants) | 2779 | 2774
  HR-HPV M24 | 2 | 6
  HPV-16 M48: number analyzed (Participants) | 2705 | 2707
  HPV-16 M48 | 1 | 7
  HPV-18 M48: number analyzed (Participants) | 2766 | 2765
  HPV-18 M48 | 0 | 0
  HPV-31 M48: number analyzed (Participants) | 2772 | 2767
  HPV-31 M48 | 0 | 2
  HPV-33 M48: number analyzed (Participants) | 2765 | 2768
  HPV-33 M48 | 1 | 2
  HPV-35 M48: number analyzed (Participants) | 2791 | 2788
  HPV-35 M48 | 0 | 2
  HPV-39 M48: number analyzed (Participants) | 2743 | 2757
  HPV-39 M48 | 1 | 0
  HPV-45 M48: number analyzed (Participants) | 2779 | 2786
  HPV-45 M48 | 0 | 0
  HPV-51 M48: number analyzed (Participants) | 2739 | 2741
  HPV-51 M48 | 0 | 0
  HPV-52 M48: number analyzed (Participants) | 2651 | 2649
  HPV-52 M48 | 2 | 1
  HPV-56 M48: number analyzed (Participants) | 2768 | 2765
  HPV-56 M48 | 0 | 0
  HPV-58 M48: number analyzed (Participants) | 2757 | 2753
  HPV-58 M48 | 4 | 2
  HPV-59 M48: number analyzed (Participants) | 2799 | 2781
  HPV-59 M48 | 0 | 0
  HPV-66 M48: number analyzed (Participants) | 2765 | 2750
  HPV-66 M48 | 2 | 1
  HPV-68 M48: number analyzed (Participants) | 2760 | 2769
  HPV-68 M48 | 0 | 0
  HPV-31/33/45 M48: number analyzed (Participants) | 2808 | 2808
  HPV-31/33/45 M48 | 1 | 4
  HPV-16/18/31/33/45 M48: number analyzed (Participants) | 2808 | 2809
  HPV-16/18/31/33/45 M48 | 2 | 11
  HRW-HPV M48: number analyzed (Participants) | 2808 | 2809
  HRW-HPV M48 | 8 | 9
  HR-HPV M48: number analyzed (Participants) | 2808 | 2809
  HR-HPV M48 | 8 | 15
  HPV-16 M57: number analyzed (Participants) | 2707 | 2710
  HPV-16 M57 | 1 | 10
  HPV-18 M57: number analyzed (Participants) | 2768 | 2768
  HPV-18 M57 | 0 | 0
  HPV-31 M57: number analyzed (Participants) | 2774 | 2770
  HPV-31 M57 | 0 | 4
  HPV-33 M57: number analyzed (Participants) | 2767 | 2771
  HPV-33 M57 | 1 | 2
  HPV-35 M57: number analyzed (Participants) | 2793 | 2791
  HPV-35 M57 | 1 | 2
  HPV-39 M57: number analyzed (Participants) | 2745 | 2760
  HPV-39 M57 | 2 | 0
  HPV-45 M57: number analyzed (Participants) | 2781 | 2789
  HPV-45 M57 | 0 | 2
  HPV-51 M57: number analyzed (Participants) | 2741 | 2743
  HPV-51 M57 | 0 | 0
  HPV-52 M57: number analyzed (Participants) | 2653 | 2652
  HPV-52 M57 | 2 | 2
  HPV-56 M57: number analyzed (Participants) | 2770 | 2767
  HPV-56 M57 | 0 | 1
  HPV-58 M57: number analyzed (Participants) | 2759 | 2756
  HPV-58 M57 | 4 | 5
  HPV-59 M57: number analyzed (Participants) | 2801 | 2784
  HPV-59 M57 | 0 | 0
  HPV-66 M57: number analyzed (Participants) | 2767 | 2752
  HPV-66 M57 | 2 | 1
  HPV-68 M57: number analyzed (Participants) | 2762 | 2772
  HPV-68 M57 | 0 | 0
  HPV-31/33/45 M57: number analyzed (Participants) | 2810 | 2811
  HPV-31/33/45 M57 | 1 | 7
  HPV-16/18/31/33/45 M57 | 2 | 17
  HRW-HPV M57 | 10 | 16
  HR-HPV M57 | 10 | 25
  HPV-16 M72: number analyzed (Participants) | 2706 | 2709
  HPV-16 M72 | 1 | 10
  HPV-18 M72: number analyzed (Participants) | 2767 | 2767
  HPV-18 M72 | 0 | 0
  HPV-31 M72: number analyzed (Participants) | 2773 | 2769
  HPV-31 M72 | 0 | 4
  HPV-33 M72: number analyzed (Participants) | 2766 | 2770
  HPV-33 M72 | 2 | 3
  HPV-35 M72: number analyzed (Participants) | 2792 | 2790
  HPV-35 M72 | 1 | 2
  HPV-39 M72: number analyzed (Participants) | 2744 | 2759
  HPV-39 M72 | 2 | 0
  HPV-45 M72: number analyzed (Participants) | 2780 | 2788
  HPV-45 M72 | 0 | 2
  HPV-51 M72: number analyzed (Participants) | 2740 | 2742
  HPV-51 M72 | 1 | 0
  HPV-52 M72: number analyzed (Participants) | 2652 | 2651
  HPV-52 M72 | 2 | 2
  HPV-56 M72: number analyzed (Participants) | 2769 | 2766
  HPV-56 M72 | 0 | 1
  HPV-58 M72: number analyzed (Participants) | 2758 | 2755
  HPV-58 M72 | 5 | 5
  HPV-59 M72: number analyzed (Participants) | 2800 | 2783
  HPV-59 M72 | 0 | 0
  HPV-66 M72: number analyzed (Participants) | 2766 | 2751
  HPV-66 M72 | 2 | 1
  HPV-68 M72: number analyzed (Participants) | 2761 | 2771
  HPV-68 M72 | 0 | 0
  HPV-31/33/45 M72: number analyzed (Participants) | 2809 | 2810
  HPV-31/33/45 M72 | 2 | 8
  HPV-16/18/31/33/45 M72: number analyzed (Participants) | 2809 | 2811
  HPV-16/18/31/33/45 M72 | 3 | 18
  HRW-HPV M72: number analyzed (Participants) | 2809 | 2811
  HRW-HPV M72 | 13 | 17
  HR-HPV M72: number analyzed (Participants) | 2809 | 2811
  HR-HPV M72 | 13 | 26

17. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Symptoms
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = solicited local symptom reported irrespective of intensity grade, Grade 3 Pain = pain that prevented normal activity, Grade 3 Swelling or Redness = swelling or redness above (>) 50 millimeter (mm). All local symptoms were considered as related to the study vaccination.
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 3005 | 3001
Participants
  Any Pain - Dose 1 | 2439 | 1815
  Grade 3 Pain - Dose 1 | 105 | 23
  Any Pain - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Pain - Dose 2 | 1650 | 1062
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Pain - Dose 2 | 53 | 17
  Any Pain - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Pain - Dose 3 | 1499 | 918
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Pain - Dose 3 | 86 | 26
  Any Pain - Across doses | 2634 | 2166
  Grade 3 Pain - Across doses | 211 | 64
  Any Redness - Dose 1 | 512 | 326
  Grade 3 Redness - Dose 1 | 1 | 1
  Any Redness - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Redness - Dose 2 | 350 | 182
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Redness - Dose 2 | 2 | 0
  Any Redness - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Redness - Dose 3 | 432 | 173
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Redness - Dose 3 | 2 | 0
  Any Redness - Across Doses | 838 | 517
  Grade 3 Redness - Across Doses | 5 | 1
  Any Swelling - Dose 1 | 514 | 215
  Grade 3 Swelling - Dose 1 | 34 | 4
  Any Swelling - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Swelling - Dose 2 | 323 | 120
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Swelling - Dose 2 | 19 | 2
  Any Swelling - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Swelling - Dose 3 | 447 | 149
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Swelling - Dose 3 | 10 | 1
  Any Swelling - Across Doses | 853 | 408
  Grade 3 Swelling - Across Doses | 48 | 5

18. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Symptoms, for Subjects Seronegative and DNA Negative for Both HPV-16 and HPV-18 at Baseline
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = solicited local symptom reported irrespective of intensity grade Grade 3 Pain = pain that prevented normal activity Grade 3 Swelling or Redness = swelling/redness above (>) 50 millimeter (mm). All local symptoms were considered as related to the study vaccination.
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1879 | 1831
Participants
  Any Pain - Dose 1 | 1519 | 1079
  Grade 3 Pain - Dose 1 | 65 | 11
  Any Pain - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Pain - Dose 2 | 1029 | 627
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Pain - Dose 2 | 35 | 10
  Any Pain - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Pain - Dose 3 | 923 | 530
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Pain - Dose 3 | 54 | 14
  Any Pain - Across doses | 1633 | 1286
  Grade 3 Pain - Across doses | 131 | 22
  Any Redness - Dose 1 | 290 | 174
  Grade 3 Redness - Dose 1 | 1 | 1
  Any Redness - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Redness - Dose 2 | 201 | 99
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Redness - Dose 2 | 0 | 0
  Any Redness - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Redness - Dose 3 | 240 | 95
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Redness - Dose 3 | 0 | 0
  Any Redness - Across doses | 486 | 280
  Grade 3 Redness - Across doses | 1 | 1
  Any Swelling - Dose 1 | 293 | 138
  Grade 3 Swelling - Dose 1 | 18 | 4
  Any Swelling - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Swelling - Dose 2 | 196 | 65
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Swelling - Dose 2 | 12 | 1
  Any Swelling - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Swelling - Dose 3 | 248 | 85
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Swelling - Dose 3 | 7 | 1
  Any Swelling - Across doses | 493 | 228
  Grade 3 Swelling - Across doses | 28 | 4

19. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Symptoms, for Subjects Seropositive and/or DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = solicited local symptom reported irrespective of intensity grade Grade 3 Pain = pain that prevented normal activity, Grade 3 Swelling or Redness = swelling/redness above (>) 50 millimeter (mm). All local symptoms were considered as related to the study vaccination.
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1124 | 1167
Participants
  Any Pain - Dose 1 | 919 | 733
  Grade 3 Pain - Dose 1 | 40 | 11
  Any Pain - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Pain - Dose 2 | 620 | 434
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Pain - Dose 2 | 18 | 7
  Any Pain - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Pain - Dose 3 | 576 | 386
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Pain - Dose 3 | 32 | 12
  Any Pain - Across doses | 1000 | 877
  Grade 3 Pain - Across doses | 80 | 30
  Any Redness - Dose 1 | 222 | 151
  Grade 3 Redness - Dose 1 | 0 | 0
  Any Redness - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Redness - Dose 2 | 148 | 83
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Redness - Dose 2 | 2 | 0
  Any Redness - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Redness - Dose 3 | 192 | 78
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Redness - Dose 3 | 2 | 0
  Any Redness - Across doses | 351 | 236
  Grade 3 Redness - Across doses | 4 | 0
  Any Swelling - Dose 1 | 220 | 112
  Grade 3 Swelling - Dose 1 | 16 | 0
  Any Swelling - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Swelling - Dose 2 | 126 | 55
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Swelling - Dose 2 | 7 | 1
  Any Swelling - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Swelling - Dose 3 | 199 | 64
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Swelling - Dose 3 | 3 | 0
  Any Swelling - Across doses | 359 | 179
  Grade 3 Swelling - Across doses | 20 | 1

20. Secondary Outcome: Number of Subjects With Any and Severe (Grade 3) Solicited Local Symptoms, for Subjects DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: Solicited local symptoms assessed were pain, redness and swelling. Any = solicited local symptom reported irrespective of intensity grade, Grade 3 Redness, Swelling = redness/swelling above 50 millimeter All local symptoms were considered as related to the study vaccination
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 151 | 127
Participants
  Any Pain - Dose 1 | 123 | 82
  Grade 3 Pain - Dose 1 | 5 | 0
  Any Pain - Dose 2: number analyzed (Participants) | 151 | 125
  Any Pain - Dose 2 | 78 | 55
  Grade 3 Pain - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Pain - Dose 2 | 2 | 1
  Any Pain - Dose 3: number analyzed (Participants) | 148 | 123
  Any Pain - Dose 3 | 74 | 43
  Grade 3 Pain - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Pain - Dose 3 | 5 | 1
  Any Pain - Across doses | 133 | 97
  Grade 3 Pain - Across doses | 11 | 3
  Any Redness - Dose 1 | 41 | 16
  Grade 3 Redness - Dose 1 | 0 | 0
  Any Redness - Dose 2: number analyzed (Participants) | 151 | 125
  Any Redness - Dose 2 | 24 | 11
  Grade 3 Redness - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Redness - Dose 2 | 0 | 0
  Any Redness - Dose 3: number analyzed (Participants) | 148 | 123
  Any Redness - Dose 3 | 23 | 6
  Grade 3 Redness - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Redness - Dose 3 | 0 | 0
  Any Redness - Across doses | 55 | 28
  Grade 3 Redness - Across doses | 0 | 0
  Any Swelling - Dose 1 | 40 | 14
  Grade 3 Swelling - Dose 1 | 0 | 0
  Any Swelling - Dose 2: number analyzed (Participants) | 151 | 125
  Any Swelling - Dose 2 | 21 | 8
  Grade 3 Swelling - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Swelling - Dose 2 | 0 | 0
  Any Swelling - Dose 3: number analyzed (Participants) | 148 | 123
  Any Swelling - Dose 3 | 29 | 5
  Grade 3 Swelling - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Swelling - Dose 3 | 0 | 0
  Any Swelling - Across doses | 58 | 21
  Grade 3 Swelling - Across doses | 0 | 0

21. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Causally Related to Vaccination Solicited General Symptoms.
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, fever (= axillary temperature above 37.0 degrees Celsius) and urticaria. Any = any solicited general symptom reported irrespective of intensity grade and relationship to vaccination, Related = symptoms assessed by the investigator as causally related to study vaccination, Grade 3 symptoms = prevented normal activity, Grade 3 urticaria = distributed on at least 4 body areas.
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 3005 | 3001
Participants
  Any Arthralgia - Dose 1 | 199 | 163
  Any Arthralgia - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Arthralgia - Dose 2 | 63 | 51
  Any Arthralgia - Dose 3: number analyzed (Participants) | 2983 | 2987
  Any Arthralgia - Dose 3 | 67 | 32
  Any Arthralgia - Across doses | 270 | 213
  Grade 3 Arthralgia - Dose 1 | 0 | 3
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Arthralgia - Dose 2 | 1 | 0
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Arthralgia - Dose 3 | 1 | 1
  Grade 3 Arthralgia - Across doses | 2 | 4
  Related Arthralgia - Dose 1 | 143 | 109
  Related Arthralgia - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Arthralgia - Dose 2 | 51 | 32
  Related Arthralgia - Dose 3: number analyzed (Participants) | 2934 | 2851
  Related Arthralgia - Dose 3 | 61 | 26
  Related Arthralgia - Across doses | 210 | 149
  Any Fatigue - Dose 1 | 817 | 769
  Any Fatigue - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Fatigue - Dose 2 | 447 | 367
  Any Fatigue - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Fatigue - Dose 3 | 443 | 309
  Any Fatigue - Across doses | 1142 | 1018
  Grade 3 Fatigue - Dose 1 | 14 | 18
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Fatigue - Dose 2 | 1 | 0
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Fatigue - Dose 3 | 5 | 5
  Grade 3 Fatigue - Across doses | 26 | 29
  Related Fatigue - Dose 1 | 634 | 581
  Related Fatigue - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Fatigue - Dose 2 | 51 | 32
  Related Fatigue - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Fatigue - Dose 3 | 390 | 256
  Related Fatigue - Across doses | 968 | 833
  Any Gastrointestinal - Dose 1 | 295 | 368
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Gastrointestinal - Dose 2 | 123 | 111
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Gastrointestinal - Dose 3 | 64 | 61
  Any Gastrointestinal - Across doses | 409 | 473
  Grade 3 Gastrointestinal - Dose 1 | 10 | 18
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Gastrointestinal - Dose 2 | 2 | 5
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Gastrointestinal - Dose 3 | 3 | 1
  Grade 3 Gastrointestinal - Across doses | 15 | 22
  Related Gastrointestinal - Dose 1 | 177 | 200
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Gastrointestinal - Dose 2 | 79 | 65
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Gastrointestinal - Dose 3 | 50 | 43
  Related Gastrointestinal - Across doses | 267 | 275
  Any Headache - Dose 1 | 476 | 509
  Any Headache - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Headache - Dose 2 | 229 | 208
  Any Headache - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Headache - Dose 3 | 191 | 146
  Any Headache - Across doses | 684 | 682
  Grade 3 Headache - Dose 1 | 332 | 347
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Headache - Dose 2 | 5 | 4
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Headache - Dose 3 | 6 | 5
  Grade 3 Headache - Across doses | 25 | 20
  Related Headache - Dose 1 | 332 | 347
  Related Headache - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Headache - Dose 2 | 180 | 161
  Related Headache - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Headache - Dose 3 | 164 | 107
  Related Headache - Across doses | 526 | 505
  Any Myalgia - Dose 1 | 362 | 249
  Any Myalgia - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Myalgia - Dose 2 | 118 | 73
  Any Myalgia - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Myalgia - Dose 3 | 175 | 109
  Any Myalgia - Across doses | 523 | 360
  Grade 3 Myalgia - Dose 1 | 5 | 2
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Myalgia - Dose 2 | 2 | 1
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Myalgia - Dose 3 | 2 | 3
  Grade 3 Myalgia - Across doses | 9 | 5
  Related Myalgia - Dose 1 | 303 | 188
  Related Myalgia - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Myalgia - Dose 2 | 98 | 57
  Related Myalgia - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Myalgia - Dose 3 | 153 | 92
  Related Myalgia - Across doses | 449 | 287
  Any Rash - Dose 1 | 28 | 42
  Any Rash - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Rash - Dose 2 | 9 | 13
  Any Rash - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Rash - Dose 3 | 12 | 7
  Any Rash - Across doses | 47 | 59
  Grade 3 Rash - Dose 1 | 1 | 1
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Rash - Dose 2 | 0 | 0
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Rash - Dose 3 | 2 | 1
  Grade 3 Rash - Across doses | 3 | 2
  Related Rash - Dose 1 | 15 | 19
  Related Rash - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Rash - Dose 2 | 1 | 9
  Related Rash - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Rash - Dose 3 | 5 | 5
  Related Rash - Across doses | 21 | 33
  >37.0°C Fever - Dose 1 | 480 | 433
  >37.0°C Fever - Dose 2: number analyzed (Participants) | 2983 | 2987
  >37.0°C Fever - Dose 2 | 232 | 236
  >37.0°C Fever - Dose 3: number analyzed (Participants) | 2934 | 2951
  >37.0°C Fever - Dose 3 | 182 | 175
  >37.0°C Fever - Across doses | 744 | 697
  >39.0°C Fever - Dose 1 | 2 | 0
  >39.0°C Fever - Dose 2: number analyzed (Participants) | 2983 | 2987
  >39.0°C Fever - Dose 2 | 6 | 0
  >39.0°C Fever - Dose 3: number analyzed (Participants) | 2934 | 2951
  >39.0°C Fever - Dose 3 | 3 | 2
  >39.0°C Fever - Across doses | 11 | 2
  Related Fever - Dose 1 | 386 | 344
  Related Fever - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Fever - Dose 2 | 175 | 168
  Related Fever - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Fever - Dose 3 | 124 | 117
  Related Fever - Across doses | 588 | 539
  Any Urticaria - Dose 1 | 22 | 20
  Any Urticaria - Dose 2: number analyzed (Participants) | 2983 | 2987
  Any Urticaria - Dose 2 | 6 | 6
  Any Urticaria - Dose 3: number analyzed (Participants) | 2934 | 2951
  Any Urticaria - Dose 3 | 4 | 4
  Any Urticaria - Across doses | 29 | 28
  Grade 3 Urticaria - Dose 1 | 4 | 2
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 2983 | 2987
  Grade 3 Urticaria - Dose 2 | 0 | 0
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 2934 | 2951
  Grade 3 Urticaria - Dose 3 | 1 | 1
  Grade 3 Urticaria - Across doses | 5 | 3
  Related Urticaria - Dose 1 | 10 | 12
  Related Urticaria - Dose 2: number analyzed (Participants) | 2983 | 2987
  Related Urticaria - Dose 2 | 6 | 5
  Related Urticaria - Dose 3: number analyzed (Participants) | 2934 | 2951
  Related Urticaria - Dose 3 | 1 | 1
  Related Urticaria - Across doses | 16 | 16

22. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Causally Related to Vaccination Solicited General Symptoms, for Subjects Seronegative and DNA Negative for Both HPV-16 and HPV-18 at Baseline
Description: Solicited general symptoms assessed were arthralgia, fatigue, gastrointestinal, headache, myalgia, rash, fever (= axillary temperature above 37.0°C) and urticaria. Any = any solicited general symptom reported irrespective of intensity grade and relationship to vaccination Related = symptoms assessed by the investigator as causally related to study vaccination Grade 3 symptoms = symptoms that prevented normal activity Grade 3 urticaria = urticaria distributed on at least 4 body areas.
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1879 | 1831
Participants
  Any Arthralgia - Dose 1 | 124 | 96
  Any Arthralgia - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Arthralgia - Dose 2 | 33 | 34
  Any Arthralgia - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Arthralgia - Dose 3 | 40 | 18
  Any Arthralgia - Across doses | 164 | 128
  Grade 3 Arthralgia - Dose 1 | 0 | 2
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Arthralgia - Dose 2 | 0 | 0
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Arthralgia - Dose 3 | 0 | 0
  Grade 3 Arthralgia - Across doses | 0 | 2
  Related Arthralgia - Dose 1 | 89 | 62
  Related Arthralgia - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Arthralgia - Dose 2 | 29 | 20
  Related Arthralgia - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Arthralgia - Dose 3 | 37 | 16
  Related Arthralgia - Across doses | 128 | 87
  Any Fatigue - Dose 1 | 509 | 443
  Any Fatigue - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Fatigue - Dose 2 | 255 | 219
  Any Fatigue - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Fatigue - Dose 3 | 278 | 165
  Any Fatigue - Across doses | 711 | 588
  Grade 3 Fatigue - Dose 1 | 10 | 13
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Fatigue - Dose 2 | 4 | 3
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Fatigue - Dose 3 | 3 | 2
  Grade 3 Fatigue - Across doses | 16 | 18
  Related Fatigue - Dose 1 | 386 | 321
  Related Fatigue - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Fatigue - Dose 2 | 223 | 185
  Related Fatigue - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Fatigue - Dose 3 | 248 | 135
  Related Fatigue - Across doses | 592 | 471
  Any Gastrointestinal - Dose 1 | 182 | 227
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Gastrointestinal - Dose 2 | 66 | 65
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Gastrointestinal - Dose 3 | 33 | 35
  Any Gastrointestinal - Across doses | 240 | 287
  Grade 3 Gastrointestinal - Dose 1 | 5 | 9
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Gastrointestinal - Dose 2 | 0 | 3
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Gastrointestinal - Dose 3 | 1 | 0
  Grade 3 Gastrointestinal - Across doses | 6 | 10
  Related Gastrointestinal - Dose 1 | 114 | 122
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Gastrointestinal - Dose 2 | 40 | 40
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Gastrointestinal - Dose 3 | 25 | 27
  Related Gastrointestinal - Across doses | 154 | 170
  Any Headache - Dose 1 | 284 | 315
  Any Headache - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Headache - Dose 2 | 118 | 120
  Any Headache - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Headache - Dose 3 | 111 | 85
  Any Headache - Across doses | 408 | 404
  Grade 3 Headache - Dose 1 | 7 | 10
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Headache - Dose 2 | 2 | 2
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Headache - Dose 3 | 2 | 2
  Grade 3 Headache - Across doses | 11 | 12
  Related Headache - Dose 1 | 186 | 212
  Related Headache - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Headache - Dose 2 | 89 | 96
  Related Headache - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Headache - Dose 3 | 97 | 60
  Related Headache - Across doses | 300 | 298
  Any Myalgia - Dose 1 | 233 | 154
  Any Myalgia - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Myalgia - Dose 2 | 73 | 38
  Any Myalgia - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Myalgia - Dose 3 | 114 | 74
  Any Myalgia - Across doses | 328 | 214
  Grade 3 Myalgia - Dose 1 | 4 | 2
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Myalgia - Dose 2 | 0 | 1
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Myalgia - Dose 3 | 0 | 1
  Grade 3 Myalgia - Across doses | 4 | 3
  Related Myalgia - Dose 1 | 194 | 117
  Related Myalgia - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Myalgia - Dose 2 | 59 | 33
  Related Myalgia - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Myalgia - Dose 3 | 100 | 62
  Related Myalgia - Across doses | 280 | 173
  Any Rash - Dose 1 | 19 | 26
  Any Rash - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Rash - Dose 2 | 6 | 7
  Any Rash - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Rash - Dose 3 | 7 | 7
  Any Rash - Across doses | 32 | 37
  Grade 3 Rash - Dose 1 | 1 | 1
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Rash - Dose 2 | 0 | 0
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Rash - Dose 3 | 1 | 1
  Grade 3 Rash - Across doses | 2 | 2
  Related Rash - Dose 1 | 8 | 11
  Related Rash - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Rash - Dose 2 | 1 | 6
  Related Rash - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Rash - Dose 3 | 2 | 5
  Related Rash - Across doses | 11 | 22
  >37.0°C Fever - Dose 1 | 296 | 261
  >37.0°C Fever - Dose 2: number analyzed (Participants) | 1863 | 1825
  >37.0°C Fever - Dose 2 | 146 | 149
  >37.0°C Fever - Dose 3: number analyzed (Participants) | 1838 | 1806
  >37.0°C Fever - Dose 3 | 107 | 108
  >37.0°C Fever - Across doses | 464 | 427
  >39.0°C Fever - Dose 1 | 2 | 0
  >39.0°C Fever - Dose 2: number analyzed (Participants) | 1863 | 1825
  >39.0°C Fever - Dose 2 | 4 | 0
  >39.0°C Fever - Dose 3: number analyzed (Participants) | 1838 | 1806
  >39.0°C Fever - Dose 3 | 0 | 0
  >39.0°C Fever - Across doses | 6 | 0
  Related Fever - Dose 1 | 226 | 211
  Related Fever - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Fever - Dose 2 | 106 | 109
  Related Fever - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Fever - Dose 3 | 74 | 72
  Related Fever - Across doses | 355 | 333
  Any Urticaria - Dose 1 | 13 | 15
  Any Urticaria - Dose 2: number analyzed (Participants) | 1863 | 1825
  Any Urticaria - Dose 2 | 5 | 4
  Any Urticaria - Dose 3: number analyzed (Participants) | 1838 | 1806
  Any Urticaria - Dose 3 | 2 | 2
  Any Urticaria - Across doses | 18 | 19
  Grade 3 Urticaria - Dose 1 | 2 | 2
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 1863 | 1825
  Grade 3 Urticaria - Dose 2 | 0 | 0
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 1838 | 1806
  Grade 3 Urticaria - Dose 3 | 1 | 0
  Grade 3 Urticaria - Across doses | 3 | 2
  Related Urticaria - Dose 1 | 7 | 8
  Related Urticaria - Dose 2: number analyzed (Participants) | 1863 | 1825
  Related Urticaria - Dose 2 | 5 | 4
  Related Urticaria - Dose 3: number analyzed (Participants) | 1838 | 1806
  Related Urticaria - Dose 3 | 0 | 1
  Related Urticaria - Across doses | 11 | 11

23. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Causally Related to Vaccination Solicited General Symptoms, for Subjects Seropositive and/or DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 22
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1124 | 1167
Participants
  Any Arthralgia - Dose 1 | 75 | 67
  Any Arthralgia - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Arthralgia - Dose 2 | 30 | 17
  Any Arthralgia - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Arthralgia - Dose 3 | 27 | 14
  Any Arthralgia - Across doses | 106 | 85
  Grade 3 Arthralgia - Dose 1 | 0 | 1
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Arthralgia - Dose 2 | 1 | 0
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Arthralgia - Dose 3 | 1 | 1
  Grade 3 Arthralgia - Across doses | 2 | 2
  Related Arthralgia - Dose 1 | 54 | 47
  Related Arthralgia - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Arthralgia - Dose 2 | 22 | 12
  Related Arthralgia - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Arthralgia - Dose 3 | 24 | 10
  Related Arthralgia - Across doses | 82 | 62
  Any Fatigue - Dose 1 | 307 | 325
  Any Fatigue - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Fatigue - Dose 2 | 191 | 147
  Any Fatigue - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Fatigue - Dose 3 | 27 | 14
  Any Fatigue - Across doses | 430 | 429
  Grade 3 Fatigue - Dose 1 | 4 | 5
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Fatigue - Dose 2 | 5 | 3
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Fatigue - Dose 3 | 2 | 3
  Grade 3 Fatigue - Across doses | 10 | 11
  Related Fatigue - Dose 1 | 247 | 259
  Related Fatigue - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Fatigue - Dose 2 | 170 | 118
  Related Fatigue - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Fatigue - Dose 3 | 142 | 120
  Related Fatigue - Across doses | 375 | 361
  Any Gastrointestinal - Dose 1 | 112 | 140
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Gastrointestinal - Dose 2 | 57 | 46
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Gastrointestinal - Dose 3 | 31 | 26
  Any Gastrointestinal - Across doses | 168 | 185
  Grade 3 Gastrointestinal - Dose 1 | 5 | 9
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Gastrointestinal - Dose 2 | 2 | 2
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Gastrointestinal - Dose 3 | 2 | 1
  Grade 3 Gastrointestinal - Across doses | 9 | 12
  Related Gastrointestinal - Dose 1 | 62 | 78
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Gastrointestinal - Dose 2 | 39 | 25
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Gastrointestinal - Dose 3 | 25 | 16
  Related Gastrointestinal - Across doses | 112 | 105
  Any Headache - Dose 1 | 191 | 193
  Any Headache - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Headache - Dose 2 | 111 | 88
  Any Headache - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Headache - Dose 3 | 80 | 61
  Any Headache - Across doses | 275 | 277
  Grade 3 Headache - Dose 1 | 7 | 3
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Headache - Dose 2 | 3 | 2
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Headache - Dose 3 | 4 | 3
  Grade 3 Headache - Across doses | 14 | 8
  Related Headache - Dose 1 | 145 | 134
  Related Headache - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Headache - Dose 2 | 91 | 65
  Related Headache - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Headache - Dose 3 | 67 | 47
  Related Headache - Across doses | 225 | 206
  Any Myalgia - Dose 1 | 129 | 94
  Any Myalgia - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Myalgia - Dose 2 | 45 | 35
  Any Myalgia - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Myalgia - Dose 3 | 61 | 35
  Any Myalgia - Across doses | 195 | 145
  Grade 3 Myalgia - Dose 1 | 1 | 0
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Myalgia - Dose 2 | 2 | 0
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Myalgia - Dose 3 | 2 | 2
  Grade 3 Myalgia - Across doses | 5 | 2
  Related Myalgia - Dose 1 | 109 | 70
  Related Myalgia - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Myalgia - Dose 2 | 39 | 24
  Related Myalgia - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Myalgia - Dose 3 | 53 | 30
  Related Myalgia - Across doses | 169 | 113
  Any Rash - Dose 1 | 9 | 16
  Any Rash - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Rash - Dose 2 | 3 | 6
  Any Rash - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Rash - Dose 3 | 5 | 0
  Any Rash - Across doses | 15 | 22
  Grade 3 Rash - Dose 1 | 0 | 0
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Rash - Dose 2 | 0 | 0
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Rash - Dose 3 | 1 | 0
  Grade 3 Rash - Across doses | 1 | 0
  Related Rash - Dose 1 | 7 | 8
  Related Rash - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Rash - Dose 2 | 0 | 0
  Related Rash - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Rash - Dose 3 | 3 | 0
  Related Rash - Across doses | 10 | 11
  >37.0°C Fever - Dose 1 | 183 | 172
  >37.0°C Fever - Dose 2: number analyzed (Participants) | 1118 | 1159
  >37.0°C Fever - Dose 2 | 85 | 87
  >37.0°C Fever - Dose 3: number analyzed (Participants) | 1094 | 1143
  >37.0°C Fever - Dose 3 | 73 | 67
  >37.0°C Fever - Across doses | 278 | 270
  >39.0°C Fever - Dose 1 | 0 | 0
  >39.0°C Fever - Dose 2: number analyzed (Participants) | 1118 | 1159
  >39.0°C Fever - Dose 2 | 2 | 0
  >39.0°C Fever - Dose 3: number analyzed (Participants) | 1094 | 1143
  >39.0°C Fever - Dose 3 | 3 | 2
  >39.0°C Fever - Across doses | 5 | 2
  Related Fever - Dose 1 | 159 | 133
  Related Fever - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Fever - Dose 2 | 68 | 59
  Related Fever - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Fever - Dose 3 | 49 | 45
  Related Fever - Across doses | 232 | 206
  Any Urticaria - Dose 1 | 9 | 5
  Any Urticaria - Dose 2: number analyzed (Participants) | 1118 | 1159
  Any Urticaria - Dose 2 | 1 | 2
  Any Urticaria - Dose 3: number analyzed (Participants) | 1094 | 1143
  Any Urticaria - Dose 3 | 2 | 2
  Any Urticaria - Across doses | 11 | 9
  Grade 3 Urticaria - Dose 1 | 2 | 0
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 1118 | 1159
  Grade 3 Urticaria - Dose 2 | 0 | 0
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 1094 | 1143
  Grade 3 Urticaria - Dose 3 | 0 | 1
  Grade 3 Urticaria - Across doses | 2 | 1
  Related Urticaria - Dose 1 | 3 | 4
  Related Urticaria - Dose 2: number analyzed (Participants) | 1118 | 1159
  Related Urticaria - Dose 2 | 1 | 1
  Related Urticaria - Dose 3: number analyzed (Participants) | 1094 | 1143
  Related Urticaria - Dose 3 | 1 | 0
  Related Urticaria - Across doses | 5 | 5

24. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Causally Related to Vaccination Solicited General Symptoms, for Subjects DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 22
Time Frame: Within 7 days (Days 0-6) after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 151 | 127
Participants
  Any Arthralgia - Dose 1 | 12 | 8
  Any Arthralgia - Dose 2: number analyzed (Participants) | 151 | 125
  Any Arthralgia - Dose 2 | 3 | 1
  Any Arthralgia - Dose 3: number analyzed (Participants) | 148 | 123
  Any Arthralgia - Dose 3 | 1 | 1
  Any Arthralgia - Across doses | 14 | 10
  Grade 3 Arthralgia - Dose 1 | 0 | 0
  Grade 3 Arthralgia - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Arthralgia - Dose 2 | 0 | 0
  Grade 3 Arthralgia - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Arthralgia - Dose 3 | 0 | 0
  Grade 3 Arthralgia - Across doses | 0 | 0
  Related Arthralgia - Dose 1 | 7 | 5
  Related Arthralgia - Dose 2: number analyzed (Participants) | 151 | 125
  Related Arthralgia - Dose 2 | 1 | 1
  Related Arthralgia - Dose 3: number analyzed (Participants) | 148 | 123
  Related Arthralgia - Dose 3 | 1 | 0
  Related Arthralgia - Across doses | 8 | 6
  Any Fatigue - Dose 1 | 44 | 46
  Any Fatigue - Dose 2: number analyzed (Participants) | 151 | 125
  Any Fatigue - Dose 2 | 29 | 18
  Any Fatigue - Dose 3: number analyzed (Participants) | 148 | 123
  Any Fatigue - Dose 3 | 24 | 14
  Any Fatigue - Across doses | 66 | 53
  Grade 3 Fatigue - Dose 1 | 0 | 0
  Grade 3 Fatigue - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Fatigue - Dose 2 | 1 | 0
  Grade 3 Fatigue - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Fatigue - Dose 3 | 1 | 1
  Grade 3 Fatigue - Across doses | 1 | 1
  Related Fatigue - Dose 1 | 35 | 36
  Related Fatigue - Dose 2: number analyzed (Participants) | 151 | 125
  Related Fatigue - Dose 2 | 26 | 13
  Related Fatigue - Dose 3: number analyzed (Participants) | 148 | 123
  Related Fatigue - Dose 3 | 20 | 14
  Related Fatigue - Across doses | 58 | 47
  Any Gastrointestinal - Dose 1 | 14 | 20
  Any Gastrointestinal - Dose 2: number analyzed (Participants) | 151 | 125
  Any Gastrointestinal - Dose 2 | 10 | 5
  Any Gastrointestinal - Dose 3: number analyzed (Participants) | 148 | 123
  Any Gastrointestinal - Dose 3 | 3 | 1
  Any Gastrointestinal - Across doses | 22 | 24
  Grade 3 Gastrointestinal - Dose 1 | 0 | 2
  Grade 3 Gastrointestinal - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Gastrointestinal - Dose 2 | 1 | 0
  Grade 3 Gastrointestinal - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Gastrointestinal - Dose 3 | 0 | 1
  Grade 3 Gastrointestinal - Across doses | 1 | 3
  Related Gastrointestinal - Dose 1 | 7 | 8
  Related Gastrointestinal - Dose 2: number analyzed (Participants) | 151 | 125
  Related Gastrointestinal - Dose 2 | 7 | 3
  Related Gastrointestinal - Dose 3: number analyzed (Participants) | 148 | 123
  Related Gastrointestinal - Dose 3 | 2 | 1
  Related Gastrointestinal - Across doses | 14 | 12
  Any Headache - Dose 1 | 25 | 20
  Any Headache - Dose 2: number analyzed (Participants) | 151 | 125
  Any Headache - Dose 2 | 17 | 9
  Any Headache - Dose 3: number analyzed (Participants) | 148 | 123
  Any Headache - Dose 3 | 8 | 6
  Any Headache - Across doses | 36 | 31
  Grade 3 Headache - Dose 1 | 1 | 0
  Grade 3 Headache - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Headache - Dose 2 | 1 | 0
  Grade 3 Headache - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Headache - Dose 3 | 1 | 0
  Grade 3 Headache - Across doses | 3 | 0
  Related Headache - Dose 1 | 15 | 11
  Related Headache - Dose 2: number analyzed (Participants) | 151 | 125
  Related Headache - Dose 2 | 16 | 7
  Related Headache - Dose 3: number analyzed (Participants) | 148 | 123
  Related Headache - Dose 3 | 7 | 5
  Related Headache - Across doses | 29 | 22
  Any Myalgia - Dose 1 | 17 | 10
  Any Myalgia - Dose 2: number analyzed (Participants) | 151 | 125
  Any Myalgia - Dose 2 | 5 | 4
  Any Myalgia - Dose 3: number analyzed (Participants) | 148 | 123
  Any Myalgia - Dose 3 | 7 | 2
  Any Myalgia - Across doses | 25 | 15
  Grade 3 Myalgia - Dose 1 | 0 | 0
  Grade 3 Myalgia - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Myalgia - Dose 2 | 0 | 0
  Grade 3 Myalgia - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Myalgia - Dose 3 | 0 | 0
  Grade 3 Myalgia - Across doses | 0 | 0
  Related Myalgia - Dose 1 | 11 | 9
  Related Myalgia - Dose 2: number analyzed (Participants) | 151 | 125
  Related Myalgia - Dose 2 | 5 | 4
  Related Myalgia - Dose 3: number analyzed (Participants) | 148 | 123
  Related Myalgia - Dose 3 | 7 | 1
  Related Myalgia - Across doses | 19 | 13
  Any Rash - Dose 1 | 1 | 0
  Any Rash - Dose 2: number analyzed (Participants) | 151 | 125
  Any Rash - Dose 2 | 2 | 2
  Any Rash - Dose 3: number analyzed (Participants) | 148 | 123
  Any Rash - Dose 3 | 1 | 0
  Any Rash - Across doses | 4 | 2
  Grade 3 Rash - Dose 1 | 0 | 0
  Grade 3 Rash - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Rash - Dose 2 | 0 | 0
  Grade 3 Rash - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Rash - Dose 3 | 0 | 0
  Grade 3 Rash - Across doses | 0 | 0
  Related Rash - Dose 1 | 1 | 0
  Related Rash - Dose 2: number analyzed (Participants) | 151 | 125
  Related Rash - Dose 2 | 0 | 2
  Related Rash - Dose 3: number analyzed (Participants) | 148 | 123
  Related Rash - Dose 3 | 0 | 0
  Related Rash - Across doses | 1 | 2
  >37.0°C Fever - Dose 1 | 16 | 18
  >37.0°C Fever - Dose 2: number analyzed (Participants) | 151 | 125
  >37.0°C Fever - Dose 2 | 11 | 12
  >37.0°C Fever - Dose 3: number analyzed (Participants) | 148 | 123
  >37.0°C Fever - Dose 3 | 15 | 3
  >37.0°C Fever - Across doses | 32 | 26
  >39.0°C Fever - Dose 1 | 0 | 0
  >39.0°C Fever - Dose 2: number analyzed (Participants) | 151 | 125
  >39.0°C Fever - Dose 2 | 0 | 0
  >39.0°C Fever - Dose 3: number analyzed (Participants) | 148 | 123
  >39.0°C Fever - Dose 3 | 2 | 0
  >39.0°C Fever - Across doses | 2 | 0
  Related Fever - Dose 1 | 13 | 13
  Related Fever - Dose 2: number analyzed (Participants) | 151 | 125
  Related Fever - Dose 2 | 8 | 7
  Related Fever - Dose 3: number analyzed (Participants) | 148 | 123
  Related Fever - Dose 3 | 8 | 2
  Related Fever - Across doses | 23 | 18
  Any Urticaria - Dose 1 | 1 | 0
  Any Urticaria - Dose 2: number analyzed (Participants) | 151 | 125
  Any Urticaria - Dose 2 | 0 | 0
  Any Urticaria - Dose 3: number analyzed (Participants) | 148 | 123
  Any Urticaria - Dose 3 | 0 | 0
  Any Urticaria - Across doses | 1 | 0
  Grade 3 Urticaria - Dose 1 | 0 | 0
  Grade 3 Urticaria - Dose 2: number analyzed (Participants) | 151 | 125
  Grade 3 Urticaria - Dose 2 | 0 | 0
  Grade 3 Urticaria - Dose 3: number analyzed (Participants) | 148 | 123
  Grade 3 Urticaria - Dose 3 | 0 | 0
  Grade 3 Urticaria - Across doses | 0 | 0
  Related Urticaria - Dose 1 | 0 | 0
  Related Urticaria - Dose 2: number analyzed (Participants) | 151 | 125
  Related Urticaria - Dose 2 | 0 | 0
  Related Urticaria - Dose 3: number analyzed (Participants) | 148 | 123
  Related Urticaria - Dose 3 | 0 | 0
  Related Urticaria - Across doses | 0 | 0

25. Secondary Outcome: Number of Subjects With Any, Severe (Grade 3) and Causally Related to Vaccination Unsolicited Adverse Events (AEs)
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Related = event assessed by the investigator as causally related to study vaccination Grade 3 = event that prevented normal activity
Time Frame: Within Days 0-29 after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 3026 | 3025
Participants
  Any AEs | 793 | 775
  Grade 3 AEs | 18 | 18
  Related AEs | 35 | 32

26. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events for Subjects Seronegative and DNA Negative for Both HPV-16 and HPV-18 at Baseline
Description: An unsolicited adverse event is any adverse event (i.e. any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product) reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within Days 0-29 after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1892 | 1843
Participants | 497 | 468

27. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events for Subjects Seropositive and/or DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 26
Time Frame: Within Days 0-29 after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1131 | 1179
Participants | 295 | 307

28. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events for Subjects DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 26
Time Frame: Within Days 0-29 after vaccination
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 151 | 128
Participants | 32 | 40

29. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that results in death, are life threatening, require hospitalization or prolongation of hospitalization, results in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subjects.
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 3026 | 3025
Participants | 56 | 81

30. Secondary Outcome: Number of Subjects With Medically Significant Conditions (MSC) Regardless of Causal Relationship to Vaccination and Intensity
Description: Medically significant conditions were defined as: adverse events (AEs) prompting emergency room or physician visits that were not (1) related to common diseases or (2) routine visits for physical examination or vaccination, or SAEs that were not related to common diseases. Common diseases included: upper respiratory infections, sinusitis, pharyngitis, gastroenteritis, urinary tract infections, cervicovaginal yeast infections, menstrual cycle abnormalities and injury.
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 3026 | 3025
Participants | 186 | 185

31. Secondary Outcome: Number of Subjects With Medically Significant Conditions Regardless of Causal Relationship to Vaccination and Intensity for Subjects Seronegative and DNA Negative for Both HPV-16 and HPV-18 at Baseline
Description: as for outcome 30
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1892 | 1843
Participants | 122 | 110

32. Secondary Outcome: Number of Subjects With Medically Significant Conditions Regardless of Causal Relationship to Vaccination and Intensity for Subjects Seropositive and/or DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 30
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 1131 | 1179
Participants | 64 | 75

33. Secondary Outcome: Number of Subjects With Medically Significant Conditions Regardless of Causal Relationship to Vaccination and Intensity for Subjects DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 30
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 151 | 128
Participants | 10 | 9

34. Secondary Outcome: Number of Subjects With Pregnancies and Outcomes of Reported Pregnancies
Description: Outcomes of pregnancies were Live infant NO apparent congenital anomaly (ACA), Live infant CA, Elective termination NO ACA, Elective termination CA, Ectopic pregnancy, Spontaneous abortion NO ACA, Stillbirth NO ACA, Stillbirth CA, Lost to follow up and Pregnancy ongoing.
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 837 | 853
Participants
  Live infant NO ACA | 648 | 657
  Live infant CA | 5 | 0
  Elective termination NO ACA | 139 | 158
  Elective termination CA | 1 | 2
  Ectopic pregnancy | 7 | 7
  Spontaneous abortion NO ACA | 16 | 13
  Stillbirth NO ACA | 0 | 2
  Stillbirth CA | 0 | 1
  Lost to follow up | 20 | 13
  Pregnancy ongoing | 1 | 0

35. Secondary Outcome: Number of Subjects With Pregnancies and Outcomes of Reported Pregnancies for Subjects Seronegative and DNA Negative for Both HPV-16 and HPV-18 at Baseline
Description: Outcomes of pregnancies were Live infant NO apparent congenital anomaly (ACA), Live infant CA, Elective termination NO ACA, Elective termination CA, Ectopic pregnancy, Spontaneous abortion NO ACA, Stillbirth NO ACA, Stillbirth CA, Lost to follow up, Pregnancy ongoing and MIssing.
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 555 | 529
Participants
  Live infant NO ACA | 436 | 411
  Live infant CA | 5 | 0
  Elective termination NO ACA | 87 | 97
  Elective termination CA | 0 | 0
  Ectopic pregnancy | 2 | 3
  Spontaneous abortion NO ACA | 10 | 8
  Spontaneous abortion CA [Month 24] | 0 | 0
  Stillbirth NO ACA | 0 | 1
  Stillbirth CA | 0 | 0
  Lost to follow up | 14 | 9
  Pregnancy ongoing | 1 | 0
  Missing | 0 | 0

36. Secondary Outcome: Number of Subjects With Pregnancies and Outcomes of Reported Pregnancies Seropositive and/or DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 35
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 282 | 324
Participants
  Live infant NO ACA | 212 | 246
  Live infant CA | 0 | 0
  Elective termination NO ACA | 52 | 61
  Elective termination CA | 1 | 2
  Ectopic pregnancy | 5 | 4
  Spontaneous abortion NO ACA | 6 | 5
  Stillbirth NO ACA | 0 | 1
  Stillbirth CA | 0 | 1
  Lost to follow up | 6 | 4
  Pregnancy ongoing | 0 | 0
  Missing | 0 | 0

37. Secondary Outcome: Number of Subjects With Pregnancies and Outcomes of Reported Pregnancies for Subjects DNA Positive for Either HPV-16 or HPV-18 at Baseline
Description: as for outcome 34
Time Frame: From Day 0 to Month 72
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 40 | 39
Participants
  Live infant NO ACA | 29 | 26
  Live infant CA | 0 | 0
  Elective termination NO ACA | 6 | 12
  Elective termination CA | 1 | 0
  Ectopic pregnancy | 3 | 1
  Spontaneous abortion NO ACA | 0 | 0
  Stillbirth NO ACA | 0 | 0
  Stillbirth CA | 0 | 0
  Lost to follow up | 1 | 0
  Pregnancy ongoing | 0 | 0
  Missing | 0 | 0

38. Secondary Outcome: Number of Subjects With HPV-16 Antibody Concentration Equal to or Above the Assay Cut-off Value, by Pre-vaccination Status
Description: HPV-16 assay cut-off value was defined as greater than or equal to (≥) 8 ELISA units per millilitre (EL.U/mL) at PRE vaccination, Month 7, 12 and 24 and ≥ 19 EL.U/mL at Month 36, 48 and 72. Seronegative (Sero-) subjects are subjects who had an antibody concentration below 8 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration ≥ 8 EL.U/mL prior to vaccination.
Time Frame: at Months 0 (PRE), 7, 12, 24, 36, 48 and 72
Population: The analysis was performed on the ATP cohort for analysis of immunogenicity, which included all evaluable subjects in the immunogenicity subset for whom data concerning immunogenicity endpoint measures were available at the specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 236 | 220
Participants
  ≥8 EL.U/mL, sero- [pre-vaccination] | 0 | 0
  ≥8 EL.U/mL, sero+ [pre-vaccination]: number analyzed (Participants) | 103 | 105
  ≥8 EL.U/mL, sero+ [pre-vaccination] | 103 | 105
  ≥8 EL.U/mL, sero- [Month 7] | 236 | 17
  ≥8 EL.U/mL, sero+ [Month 7]: number analyzed (Participants) | 103 | 105
  ≥8 EL.U/mL, sero+ [Month 7] | 103 | 97
  ≥8 EL.U/mL, sero-, [Month12]: number analyzed (Participants) | 222 | 212
  ≥8 EL.U/mL, sero-, [Month12] | 222 | 39
  ≥8 EL.U/mL, sero+, [Month12]: number analyzed (Participants) | 99 | 97
  ≥8 EL.U/mL, sero+, [Month12] | 99 | 93
  ≥8 EL.U/mL, sero-, [Month24]: number analyzed (Participants) | 207 | 197
  ≥8 EL.U/mL, sero-, [Month24] | 207 | 31
  ≥8 EL.U/mL, sero+, [Month24]: number analyzed (Participants) | 94 | 93
  ≥8 EL.U/mL, sero+, [Month24] | 94 | 85
  ≥19 EL.U/mL, sero-, [Month 36]: number analyzed (Participants) | 183 | 162
  ≥19 EL.U/mL, sero-, [Month 36] | 183 | 4
  ≥19 EL.U/mL, sero+, [Month 36]: number analyzed (Participants) | 76 | 81
  ≥19 EL.U/mL, sero+, [Month 36] | 76 | 44
  ≥19 EL.U/mL, sero-, [Month 48]: number analyzed (Participants) | 197 | 174
  ≥19 EL.U/mL, sero-, [Month 48] | 195 | 12
  ≥19 EL.U/mL, sero+, [Month 48]: number analyzed (Participants) | 84 | 84
  ≥19 EL.U/mL, sero+, [Month 48] | 83 | 48
  ≥19 EL.U/mL, sero-, [Month 72]: number analyzed (Participants) | 160 | 164
  ≥19 EL.U/mL, sero-, [Month 72] | 153 | 10
  ≥19 EL.U/mL, sero+, [Month 72]: number analyzed (Participants) | 69 | 72
  ≥19 EL.U/mL, sero+, [Month 72] | 65 | 22

39. Secondary Outcome: Number of Subjects With HPV-18 Antibody Concentration Equal to or Above the Assay Cut-off Value, by Pre-vaccination Status
Description: HPV-18 assay cut-off value was defined as ≥ 7 EL.U/mL at PRE vaccination, Month 7, 12 and 24 and ≥ 18 EL.U/mL at Month 36, 48 and 72. Seronegative (Sero-) subjects are subjects who had an antibody concentration below 7 EL.U/mL and 18 EL.U/mL prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration ≥ 7 EL.U/mL and 18 EL.U/mL prior to vaccination.
Time Frame: at Months 0 (PRE), 7, 12, 24, 36, 48 and 72
Population: as for outcome 38
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 279 | 278
Participants
  ≥ 7 EL.U/mL, sero- PRE | 0 | 0
  ≥ 7 EL.U/mL, sero+ PRE: number analyzed (Participants) | 60 | 47
  ≥ 7 EL.U/mL, sero+ PRE | 60 | 47
  ≥ 7 EL.U/mL, sero- [Month 7] | 278 | 14
  ≥ 7 EL.U/mL, sero+ [Month 7]: number analyzed (Participants) | 60 | 47
  ≥ 7 EL.U/mL, sero+ [Month 7] | 60 | 39
  ≥ 7 EL.U/mL, sero- [Month 12]: number analyzed (Participants) | 264 | 267
  ≥ 7 EL.U/mL, sero- [Month 12] | 263 | 34
  ≥ 7 EL.U/mL, sero+ [Month 12]: number analyzed (Participants) | 57 | 42
  ≥ 7 EL.U/mL, sero+ [Month 12] | 57 | 32
  ≥ 7 EL.U/mL, sero- [Month 24]: number analyzed (Participants) | 250 | 250
  ≥ 7 EL.U/mL, sero- [Month 24] | 249 | 63
  ≥ 7 EL.U/mL, sero+ [Month 24]: number analyzed (Participants) | 51 | 40
  ≥ 7 EL.U/mL, sero+ [Month 24] | 51 | 33
  ≥ 18 EL.U/mL, sero- [Month 36]: number analyzed (Participants) | 218 | 209
  ≥ 18 EL.U/mL, sero- [Month 36] | 218 | 13
  ≥ 18 EL.U/mL, sero+ [Month 36]: number analyzed (Participants) | 41 | 34
  ≥ 18 EL.U/mL, sero+ [Month 36] | 41 | 22
  ≥ 18 EL.U/mL, sero- [Month 48]: number analyzed (Participants) | 234 | 221
  ≥ 18 EL.U/mL, sero- [Month 48] | 231 | 14
  ≥ 18 EL.U/mL, sero+ [Month 48]: number analyzed (Participants) | 47 | 37
  ≥ 18 EL.U/mL, sero+ [Month 48] | 47 | 23
  ≥ 18 EL.U/mL, sero- [Month 72]: number analyzed (Participants) | 191 | 205
  ≥ 18 EL.U/mL, sero- [Month 72] | 183 | 14
  ≥ 18 EL.U/mL, sero+ [Month 72]: number analyzed (Participants) | 38 | 31
  ≥ 18 EL.U/mL, sero+ [Month 72] | 37 | 19

40. Secondary Outcome: Geometric Mean Titers for HPV-16/HPV-18 Antibodies, by Pre-vaccination Status
Description: Titers were expressed as geometric mean titers calculated on all subjects, HPV-16 assay cut-off value was defined as greater than or equal to 8 EL.U/mL at Months 0, 7, 12 and 24 and greater than or equal to 19 EL.U/mL at Months 36, 48 and 72. HPV-18 assay cut-off value was defined as ≥ 7 EL.U/mL at Month 0, 7, 12 and 24 and ≥ 18 EL.U/mL at Months 36, 48 and 72. Seronegative (Sero-) subjects are subjects who had an antibody concentration below the assay cut-off value prior to vaccination. Seropositive (Sero+) subjects are subjects who had an antibody concentration ≥ the assay cut-off value prior to vaccination.
Time Frame: at Months 0 (PRE), 7, 12, 24, 36, 48 and 72
Population: as for outcome 38
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Cervarix Group | Placebo Group
Number analyzed (Participants) | 279 | 362
Titers
  HPV-16, sero- [pre-vaccination]: number analyzed (Participants) | 236 | 220
  HPV-16, sero- [pre-vaccination] | 4.0 [4.0 to 4.0] | 4.0 [4.0 to 4.0]
  HPV-16, sero- [Month 7]: number analyzed (Participants) | 236 | 220
  HPV-16, sero- [Month 7] | 6964.3 [6164.3 to 7868.2] | 4.6 [4.2 to 5.1]
  HPV-16, sero-, [Month 12]: number analyzed (Participants) | 222 | 212
  HPV-16, sero-, [Month 12] | 3451.3 [3055.5 to 3898.4] | 5.0 [4.7 to 5.4]
  HPV-16, sero-, [Month 24]: number analyzed (Participants) | 207 | 197
  HPV-16, sero-, [Month 24] | 1253.2 [1120.6 to 1401.5] | 4.7 [4.5 to 5.0]
  HPV-16, sero-, [Month 36]: number analyzed (Participants) | 183 | 162
  HPV-16, sero-, [Month 36] | 1074.6 [958.0 to 1205.4] | 9.8 [9.5 to 10.1]
  HPV-16, sero-, [Month 48]: number analyzed (Participants) | 197 | 174
  HPV-16, sero-, [Month 48] | 828.4 [728.4 to 942.2] | 10.7 [9.9 to 11.5]
  HPV-16, sero-, [Month 72]: number analyzed (Participants) | 160 | 164
  HPV-16, sero-, [Month 72] | 678.1 [552.9 to 831.5] | 10.5 [9.7 to 11.4]
  HPV-16, sero+ [pre-vaccination]: number analyzed (Participants) | 103 | 105
  HPV-16, sero+ [pre-vaccination] | 27.4 [22.7 to 33.0] | 25.2 [21.1 to 30.1]
  HPV-16, sero+ [Month 7]: number analyzed (Participants) | 103 | 105
  HPV-16, sero+ [Month 7] | 5672.0 [4661.9 to 6900.9] | 25.6 [20.6 to 31.9]
  HPV-16, sero+, [Month 12]: number analyzed (Participants) | 99 | 97
  HPV-16, sero+, [Month 12] | 3219.8 [2593.3 to 3997.7] | 28.5 [23.2 to 35.1]
  HPV-16, sero+, [Month 24]: number analyzed (Participants) | 94 | 93
  HPV-16, sero+, [Month 24] | 1317.7 [1094.4 to 1586.5] | 19.7 [16.1 to 24.1]
  HPV-16, sero+, [Month 36]: number analyzed (Participants) | 76 | 81
  HPV-16, sero+, [Month 36] | 1290.3 [1071.7 to 1553.5] | 24.6 [19.4 to 31.2]
  HPV-16, sero+, [Month 48]: number analyzed (Participants) | 84 | 84
  HPV-16, sero+, [Month 48] | 1006.0 [817.9 to 1237.2] | 25.1 [20.1 to 31.4]
  HPV-16, sero+, [Month 72]: number analyzed (Participants) | 69 | 72
  HPV-16, sero+, [Month 72] | 724.4 [503.1 to 1043.0] | 17.3 [13.5 to 22.3]
  HPV-18, sero- [pre-vaccination]: number analyzed (Participants) | 279 | 278
  HPV-18, sero- [pre-vaccination] | 3.5 [3.5 to 3.5] | 3.5 [3.5 to 3.5]
  HPV-18, sero- [Month 7]: number analyzed (Participants) | 279 | 278
  HPV-18, sero- [Month 7] | 3357.4 [2974.7 to 3789.4] | 3.9 [3.6 to 4.2]
  HPV-18, sero-, [Month 12]: number analyzed (Participants) | 264 | 267
  HPV-18, sero-, [Month 12] | 1318.9 [1166.2 to 1491.4] | 4.2 [4.0 to 4.5]
  HPV-18, sero-, [Month 24]: number analyzed (Participants) | 250 | 250
  HPV-18, sero-, [Month 24] | 711.7 [629.6 to 804.6] | 5.0 [4.6 to 5.4]
  HPV-18, sero-, [Month 36]: number analyzed (Participants) | 218 | 209
  HPV-18, sero-, [Month 36] | 525.1 [467.2 to 590.3] | 9.7 [9.3 to 10.1]
  HPV-18, sero-, [Month 48]: number analyzed (Participants) | 234 | 221
  HPV-18, sero-, [Month 48] | 387.7 [342.6 to 438.8] | 9.8 [9.3 to 10.3]
  HPV-18, sero-, [Month 72]: number analyzed (Participants) | 191 | 205
  HPV-18, sero-, [Month 72] | 343.7 [291.9 to 404.8] | 10.1 [9.4 to 11.0]
  HPV-18, sero+ [pre-vaccination]: number analyzed (Participants) | 60 | 47
  HPV-18, sero+ [pre-vaccination] | 19.9 [16.4 to 24.1] | 25.8 [19.5 to 34.1]
  HPV-18, sero+ [Month 7]: number analyzed (Participants) | 60 | 47
  HPV-18, sero+ [Month 7] | 3200.2 [2690.8 to 3806.1] | 24.2 [15.8 to 36.9]
  HPV-18, sero+, [Month 12]: number analyzed (Participants) | 57 | 42
  HPV-18, sero+, [Month 12] | 1152.9 [932.3 to 1425.6] | 20.2 [13.7 to 30.0]
  HPV-18, sero+, [Month 24]: number analyzed (Participants) | 51 | 40
  HPV-18, sero+, [Month 24] | 831.6 [659.5 to 1048.7] | 21.9 [15.1 to 31.8]
  HPV-18, sero+, [Month 36]: number analyzed (Participants) | 41 | 34
  HPV-18, sero+, [Month 36] | 601.8 [465.4 to 778.0] | 33.4 [22.4 to 49.8]
  HPV-18, sero+, [Month 48]: number analyzed (Participants) | 47 | 37
  HPV-18, sero+, [Month 48] | 523.0 [403.8 to 677.5] | 25.5 [18.3 to 35.4]
  HPV-18, sero+, [Month 72]: number analyzed (Participants) | 38 | 31
  HPV-18, sero+, [Month 72] | 420.0 [278.9 to 632.4] | 28.3 [19.0 to 42.1]

ADVERSE EVENTS:
Time Frame: SAEs: up to Month 72. Unsolicited AEs: Within Days 0-29 after vaccination. Solicited local and general symptoms: Within 7 days (Days 0-6) after vaccination
Description: Safety data presented here were assessed for all vaccinated subjects for whom data were available at the time of the event-triggered analysis irrespective of the initial (Month 0) HPV-16 or HPV-18 serostatus and DNA status.
Arm/Group | Cervarix Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/3026 | 3/3025
Serious Adverse Events (participants affected / at risk) | 56/3026 | 81/3025
Other Adverse Events (participants affected / at risk) | 2786/3026 | 2548/3025
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix Group (N=3026) | Placebo Group (N=3025)
Appendicitis (Infections and infestations) | 4 | 12
Ectopic pregnancy (General disorders) | 6 | 6
Abortion missed (Pregnancy, puerperium and perinatal conditions) | 5 | 3
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 5 | 3
Breast cyst (Reproductive system and breast disorders) | 1 | 1
Ectopic pregnancy with intrauterine device (General disorders) | 1 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 1 | 1
Ovarian cyst torsion (Reproductive system and breast disorders) | 1 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abortion spontaneous complete (Pregnancy, puerperium and perinatal conditions) | 2 | 5
Premature baby (Pregnancy, puerperium and perinatal conditions) | 1 | 5
Abortion induced (Surgical and medical procedures) | 1 | 2
Comminuted fracture (Injury, poisoning and procedural complications) | 0 | 3
Haemorrhage intracranial (Nervous system disorders) | 1 | 2
Ovarian cyst (Reproductive system and breast disorders) | 2 | 1
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 1 | 2
Cholelithiasis (Gastrointestinal disorders) | 0 | 2
Chronic tonsillitis (Infections and infestations) | 0 | 2
Cleft lip and palate (Congenital, familial and genetic disorders) | 2 | 0
Completed suicide (Psychiatric disorders) | 0 | 2
Concussion (Injury, poisoning and procedural complications) | 0 | 2
Congenital torticollis (Congenital, familial and genetic disorders) | 2 | 0
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 | 1
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 1 | 1
Neonatal pneumonia (Infections and infestations) | 1 | 1
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Premature separation of placenta (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 0 | 2
Teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Abdominal injury (Injury, poisoning and procedural complications) | 1 | 0
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Amputation (Surgical and medical procedures) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 1
Angiomyolipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atrial septal defect (Congenital, familial and genetic disorders) | 1 | 0
Benign gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Blighted ovum (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1
Chondrodystrophy (Congenital, familial and genetic disorders) | 1 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 | 0
Cyst (General disorders) | 0 | 1
Diaphragmatic hernia (Gastrointestinal disorders) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 0 | 1
IgA nephropathy (Renal and urinary disorders) | 1 | 0
Imminent abortion (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Iris injury (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Myocarditis (Cardiac disorders) | 0 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 1 | 0
Pelvic infection (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Placental insufficiency (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Pulmonary hypoplasia (Congenital, familial and genetic disorders) | 0 | 1
Renal disorder (Renal and urinary disorders) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Trisomy 21 (Congenital, familial and genetic disorders) | 0 | 1
Urethral cyst (Renal and urinary disorders) | 0 | 1
Uterine cyst (Reproductive system and breast disorders) | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 1 | 0
Vascular rupture (Vascular disorders) | 0 | 1
Wound (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Cervarix Group (N=3026) | Placebo Group (N=3025)
Upper respiratory tract infection (Infections and infestations) | 276 | 290
Pain (General disorders) | 2634/3005 | 2166/3001
Erythema (Skin and subcutaneous tissue disorders) | 838/3005 | 517/3001
Swelling (General disorders) | 853/3005 | 408/3001
Arthralgia (Musculoskeletal and connective tissue disorders) | 270/3005 | 213/3001
Fatigue (General disorders) | 1142/3005 | 1018/3001
Gastrointestinal (Gastrointestinal disorders) | 409/3005 | 473/3001
Headache (Nervous system disorders) | 691/3005 | 690/3001
Myalgia (Musculoskeletal and connective tissue disorders) | 523/3005 | 360/3001
Pyrexia (General disorders) | 749/3005 | 703/3001

LIMITATIONS AND CAVEATS:
At the time of the event-triggered analysis at Month 24, some safety results remain blinded and are not presented here since the study is still ongoing. These results will be updated once they become available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.